CLINICAL TRIAL: NCT02159066
Title: The LOGIC 2 Trial A Phase II, Multi-center, Open-label Study of Sequential LGX818/MEK162 Combination Followed by a Rational Combination With Targeted Agents After Progression, to Overcome Resistance in Adult Patients With Locally Advanced or Metastatic BRAF V600 Melanoma.
Brief Title: LGX818 and MEK162 in Combination With a Third Agent (BKM120, LEE011, BGJ398 or INC280) in Advanced BRAF Melanoma
Acronym: LOGIC-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLGX818X2109; C4221013 (Other: Alias Study Number); 2013-004552-38 (EudraCT Number)
Record Dates: First submitted 2014-04-28; First posted 2014-06-09 (Estimated); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Melanoma
Keywords: Melanoma
MeSH Terms: conditions — Melanoma | interventions — encorafenib; binimetinib; ribociclib; infigratinib; NVP-BKM120; capmatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- LGX818 + MEK162 (Experimental)
  Interventions: Drug: LGX818; Drug: MEK162
- LGX818 + MEK162 + LEE011 (Experimental)
  Interventions: Drug: LEE011
- LGX818 + MEK162 + BGJ398 (Experimental)
  Interventions: Drug: BGJ398
- LGX818 + MEK162 + BKM120 (Experimental)
  Interventions: Drug: BKM120
- LGX818 + MEK162 + INC280 (Experimental)
  Interventions: Drug: INC280

INTERVENTIONS:
Drug: LGX818 — Combination of LGX818 and MEK162 (Part I)
  Arms: LGX818 + MEK162
Drug: MEK162 — Combination of LGX818 and MEK162 (Part I)
  Arms: LGX818 + MEK162
Drug: LEE011 — Combination of LGX818 + MEK162 + LEE011 (Part II)
  Arms: LGX818 + MEK162 + LEE011
Drug: BGJ398 — Combination of LGX818 + MEK162 + BGJ398 (Part II)
  Arms: LGX818 + MEK162 + BGJ398
Drug: BKM120 — Combination of LGX818 + MEK162 + BKM120 (Part II)
  Arms: LGX818 + MEK162 + BKM120
Drug: INC280 — Combination of LGX818 + MEK162 + INC280 (Part II)
  Arms: LGX818 + MEK162 + INC280

SUMMARY:
The primary purpose of this study is to assess the anti-tumor activity of LGX818/MEK162 in combination with targeted agents after progression on LGX818/MEK162 combination therapy, as well as the safety and tolerability of the novel triple combinations.

DETAILED DESCRIPTION:
This study consists of two parts: in Part I/Run-In, patients naïve to selective BRAF and MEK inhibitors will be treated with the LGX818/MEK162 combination until disease progression (as defined per RECIST v1.1). Based on the genetic analysis of a tumor biopsy obtained at that time, patients will enter Part II of the study for tailored combination treatment in one of four arms of LGX818/MEK162 + either BKM120, BGJ398, INC280 or LEE011 Patients with BRAF mutant melanoma treated by LGX818/MEK162 combination in other studies can be enrolled directly in Part II of CLGX818X2109 after relapse.

Dose-escalations in the combination arms for which no MTD has been established will be based on the recommendations of a Bayesian logistic regression model guided by an escalation with overdose control criterion

ELIGIBILITY:
INCLUSION CRITERIA:

* Age ≥ 18 years
* Histologically confirmed diagnosis of unresectable stage III or metastatic melanoma (stage IIIC to IV per American Joint Committee on Cancer [AJCC])
* Documented evidence of BRAF V600 mutation.
* Newly obtained tumor biopsy at baseline, and patient agrees to a mandatory biopsy at the time of progression, if not medically contraindicated.
* Evidence of measurable disease, as determined by RECIST v1.1.

INCLUSION CRITERIA for triple combinations:

Progressive disease following prior treatment with LGX818/MEK162 combination. PRINCIPAL EXCLUSION CRITERIA Symptomatic or untreated leptomeningeal disease.

* Symptomatic brain metastases. Patients previously treated or untreated for brain metastases that are asymptomatic in the absence of corticosteroid therapy or on a stable dose of steroids for four weeks are allowed to enroll. Brain metastases must be stable at least 4 weeks with verification by imaging (e.g. brain MRI completed at screening demonstrating no current evidence of progressive brain metastases). Patients are not permitted to receive enzyme inducing anti-epileptic drugs.
* Patients who have developed brain metastases during Part I of the study may continue to Part II upon discussion with Novartis Medical Monitor. The brain metastasis must be either asymptomatic or treated and stable for at least 4 weeks and on a stable or tapering dose of steroids for at least 2 weeks. Patients with brain metastasis are not eligible for the combination with LEE011.
* Known acute or chronic pancreatitis.
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes);
* Clinically significant cardiac disease including any of the following:
* CHF requiring treatment (NYH grade ≥ 2),
* LVEF < 50% as determined by MUGA scan or ECHO
* History or presence of clinically significant ventricular arrhythmias or atrial fibrillation
* Clinically significant resting bradycardia
* Unstable angina pectoris ≤ 3 months prior to starting study drug
* Acute Myocardial Infarction (AMI) ≤ 3 months prior to starting study drug,
* QTcF > 480 msec. Patients with any of the following laboratory values at

Screening/baseline:

* Absolute neutrophil count (ANC) <1,500/mm3 [1.5 x 109/L]
* Platelets < 100,000/mm3 [100 x 109/L]
* Hemoglobin < 9.0 g/dL
* Serum creatinine >1.5 x ULN or calculated or directly measured CrCl < 50% LLN (lower limit of normal)
* Serum total bilirubin >1.5 x ULN
* AST/SGOT or ALT/SGPT > 2.5 x ULN, or > 5 x ULN if liver metastases are present

Additional exclusion criteria for the triple combinations:

LGX818/MEK162/BKM120:

* Patients with fasting glucose > 120 mg/dL or 6.7 mmol/L, and HbA1c > 8 %.
* Patient has any of the following mood disorders as judged by the

Investigator or a Psychiatrist:

* Patient has a score ≥ 12 on the PHQ-9 questionnaire
* Patient has ≥ CTCAE grade 3 anxiety

LGX818/MEK162/BGJ398:

* History and/or current evidence of significant ectopic mineralization/ calcification with the exception of calcified lymph nodes and asymptomatic vascular calcification.
* Current evidence of corneal disorder/ keratopathy incl. but not limited to bullous/ band keratopathy, corneal abrasion, inflammation/ulceration, keratoconjunctivits etc., confirmed by ophthalmologic examination

LGX818/MEK162/LEE011:

* Patients with uncontrolled hypertension (please refer to WHO-ISHguidelines) are excluded from study.
* QTcF >450 ms for males and >470 ms for females Congenital long QT syndrome or family history of unexpected sudden cardiac death and/or hypokalemia CTCAE Grade ≥ 3 and magnesium levels below the clinically relevant lower limits at study entry
* Current evidence of brain metastasis or brain metastasis detected by mandatory CT/MRI at screening
* PT/INR or aPTT > 1.5xULN

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2014-07-23 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (32):
- United States (17):
  - University of California Los Angeles, Los Angeles, California
  - Cancer Care Center, Los Angeles, California
  - Doris Stein Research Center Building, Los Angeles, California
  - Ronald Reagan UCLA Medical Center Drug Information Center Department of Pharmaceutical Services, Los Angeles, California
  - UCLA Dermatology Clinic, Los Angeles, California
  - UCLA Oncology Center, Los Angeles, California
  - UCLA Radiology, Los Angeles, California
  - Memorial Sloan Kettering Cancer Center Attn: Geny O'neill, New York, New York
  - Memorial Sloan Kettering Cancer Center Inpatient Hospital & Main Campus, New York, New York
  - Memorial Sloan Kettering Cancer Center- Outpatient Clinic, New York, New York
  - OHSU Knight Cancer Institute, Portland, Oregon
  - OHSU Center for Health and Healing 2, Portland, Oregon
  - OHSU Center for Health and Healing, Portland, Oregon
  - OHSU Research Pharmacy Services, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
- Australia (2):
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - East St Kilda Eye Clinic, Melbourne, Victoria
- Canada (2):
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Sir Mortimer B. Davis-Jewish General Hospital, Monteral, Quebec
- Germany (5):
  - University Clinic Heidelberg PPDS, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Uniklinik Köln, Cologne
  - Städtisches Klinikum München, München
  - Universitätsklinikum Würzburg, Würzburg
- Italy (2):
  - Azienda Ospedaliera Monaldi, Napoli, Campania
  - U.O.C. Oncologia Medica e Terapie Innovative Dipartimento di Melanoma IRCCS Fondazione G. Pascale, Napoli
- Het Nederlands Kanker Instituut Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam, Netherlands
- Hospital Universitario Vall d'Hebrón - PPDS, Barcelona Cataluna, Barcelona, Spain
- Universitätsspital Zürich, Zurich Flughafen, Switzerland
- Churchill Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Nassar KW, Hintzsche JD, Bagby SM, Espinoza V, Langouet-Astrie C, Amato CM, Chimed TS, Fujita M, Robinson W, Tan AC, Schweppe RE. Targeting CDK4/6 Represents a Therapeutic Vulnerability in Acquired BRAF/MEK Inhibitor-Resistant Melanoma. Mol Cancer Ther. 2021 Oct;20(10):2049-2060. doi: 10.1158/1535-7163.MCT-20-1126. Epub 2021 Aug 10. PMID 34376578

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study had 2 parts. In Part I, 158 participants were enrolled and treated with encorafenib/ binimetinib (LGX818/MEK162) combination until disease progression (PD) [as per RECISTv1.1]. Based on the genetic assessment of a tumor biopsy obtained at PD, participants from Part I entered Part II. In Part II, 58 participants received tailored combination treatment in one of the 4 arms: encorafenib/ binimetinib + buparlisib (BKM120), infigratinib (BGJ398), capmatinib (INC280) or ribociclib (LEE011).
Groups:
- Part I: Encorafenib + Binimetinib (Naive): Participants naive to selective V-raf murine sarcoma viral oncogene homolog B1 (BRAF) and mitogen-activated protein kinase (MEK) inhibitors, received encorafenib 450 milligram (mg) once a day and binimetinib 45 mg twice a day until disease progression or no clinical benefit and initiation of triple combination treatment. No dose reduction below 150 mg for encorafenib and 15 mg for binimetinib was permitted for this study. Treatment cycle for encorafenib and binimetinib was defined as 21 days of daily continuous treatment.
- Part I: Encorafenib + Binimetinib (Non-naive): Participants non-naive to selective BRAF and MEK inhibitors, received encorafenib 450 mg once a day and binimetinib 45 mg twice a day until disease progression or no clinical benefit and initiation of triple combination treatment. No dose reduction below 150 mg for encorafenib and 15 mg for binimetinib was permitted for this study. Treatment cycle for both drugs was defined as 21 days of daily continuous treatment.
- Part II: Encorafenib + Binimetinib + Ribociclib: Participants, received encorafenib 200 mg (starting dose) once a day, binimetinib 45 mg (starting dose) twice a day and ribociclib 100 mg (starting dose) once a day until disease progression or no clinical benefit. No dose reduction below 50 mg for encorafenib and 15 mg for binimetinib was permitted for this study. For ribociclib dose escalation was allowed till 600 mg and dose reduction was permitted till 50 mg. Ribociclib was taken for 21 consecutive days followed by a 7-day planned break. Treatment cycle =28 days.
- Part II: Encorafenib + Binimetinib + Infigratinib: Participants, received encorafenib 450 mg (starting dose) once a day, binimetinib 45 mg (starting dose) twice a day and infigratinib 75 mg (starting dose) once a day until disease progression or no clinical benefit. No dose reduction below 150 mg for encorafenib and 15 mg for binimetinib was permitted for this study. For infigratinib dose escalation was allowed till 125 mg and dose reduction was permitted till 25 mg. Infigratinib was taken for 21 consecutive days followed by a 7-day planned break. Treatment cycle =28 days.
- Part II: Encorafenib + Binimetinib + Capmatinib: Participants, received encorafenib 200 mg (starting dose) once a day, binimetinib 45 mg (starting dose) twice a day and capmatinib 200 mg (starting dose) capsule or 400 mg (starting dose) tablet twice a day until disease progression or no clinical benefit. No dose reduction below 50 mg for encorafenib and 15 mg for binimetinib was permitted for this study. For capmatinib dose escalation was allowed till 600 mg and dose reduction was permitted till 50 mg. Treatment cycle for encorafenib, binimetinib and capmatinib was defined as 21 days of daily continuous treatment.
- Part II: Encorafenib + Binimetinib + Buparlisib: Participants, received encorafenib 450 mg (starting dose) once a day, binimetinib 45 mg (starting dose) twice a day and buparlisib 60 mg (starting dose) once a day until disease progression or no clinical benefit. No dose reduction below 150 mg for encorafenib and 15 mg for binimetinib was permitted for this study. For buparlisib dose escalation was allowed till 100 mg and dose reduction was permitted till 30 mg. Treatment cycle for encorafenib, binimetinib and buparlisib was defined as 21 days of daily continuous treatment.
Period: Part I
Arm/Group | Part I: Encorafenib + Binimetinib (Naive) | Part I: Encorafenib + Binimetinib (Non-naive) | Part II: Encorafenib + Binimetinib + Ribociclib | Part II: Encorafenib + Binimetinib + Infigratinib | Part II: Encorafenib + Binimetinib + Capmatinib | Part II: Encorafenib + Binimetinib + Buparlisib
Started | 75 (Participants enrolled in Part I of the study.) | 83 (Participants enrolled in Part I of the study.) | 0 | 0 | 0 | 0
Completed | 0 | 4 | 0 | 0 | 0 | 0
Not Completed | 75 | 79 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 5 | 0 | 0 | 0 | 0
Not completed — Death | 11 | 9 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 37 | 46 | 0 | 0 | 0 | 0
Not completed — New Therapy for Study Indication | 5 | 4 | 0 | 0 | 0 | 0
Not completed — Termination of participants from the study | 3 | 3 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 9 | 0 | 0 | 0 | 0
Not completed — Participant/Guardian Decision | 9 | 3 | 0 | 0 | 0 | 0
Not completed — Missing Data | 1 | 0 | 0 | 0 | 0 | 0
Period: Part II
Arm/Group | Part I: Encorafenib + Binimetinib (Naive) | Part I: Encorafenib + Binimetinib (Non-naive) | Part II: Encorafenib + Binimetinib + Ribociclib | Part II: Encorafenib + Binimetinib + Infigratinib | Part II: Encorafenib + Binimetinib + Capmatinib | Part II: Encorafenib + Binimetinib + Buparlisib
Started | 0 (This reporting arm is for Part I.) | 0 (This reporting arm is for Part I.) | 38 (Eligible Part I participants enrolled in Part II to receive triple-combination.) | 1 (Eligible Part I participants enrolled in Part II to receive triple-combination.) | 13 (Eligible Part I participants enrolled in Part II to receive triple-combination.) | 6 (Eligible Part I participants enrolled in Part II to receive triple-combination.)
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 38 | 1 | 13 | 6
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 1 | 0 | 2 | 1
Not completed — Progressive Disease | 0 | 0 | 35 | 1 | 7 | 4
Not completed — New Therapy for Study Indication | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Participant/Guardian Decision | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population: participants who were treated with at least 1 dose (partial or full) of encorafenib or binimetinib in Part I and at least 1 dose of encorafenib or binimetinib or the assigned third agent following the assignment of the triple combination treatment in Part II. Parts I and II participants are not exclusive. To avoid risk of identification of participant, baseline measure data is not disclosed for reporting arm including Infigratinib and reported under category- Not Disclosed.
Groups:
- Part I: Encorafenib + Binimetinib (Naive): Participants naive to selective V-raf murine sarcoma viral oncogene homolog B1 (BRAF) and mitogen-activated protein kinase (MEK) inhibitors, received encorafenib 450 milligram (mg) once a day and binimetinib 45 mg twice a day until disease progression or no clinical benefit. No dose reduction below 150 mg for encorafenib and 15 mg for binimetinib was permitted for this study. Treatment cycle for encorafenib and binimetinib was defined as 21 days of daily continuous treatment.
- Total: Total of all reporting groups
Arm/Group | Part I: Encorafenib + Binimetinib (Naive) | Part I: Encorafenib + Binimetinib (Non-naive) | Part II: Encorafenib + Binimetinib + Ribociclib | Part II: Encorafenib + Binimetinib + Infigratinib | Part II: Encorafenib + Binimetinib + Capmatinib | Part II: Encorafenib + Binimetinib + Buparlisib | Total
Number analyzed (Participants) | 75 | 83 | 38 | 1 | 13 | 6 | 216
Age, Customized [Count of Participants; unit: Participants] — Data for arm - Part II: Encorafenib + Binimetinib + Infigratinib is not disclosed to avoid risk of identification and kept under category Not disclosed category. Population: Number Analyzed for Part I and Part II = number of participants analyzed for reporting arms for respective parts. Part I and Part II participants are not exclusive.
  Participants
    Part I: number analyzed (Participants) | 75 | 83 | 0 | 0 | 0 | 0 | 158
    Part I: 18-44 years | 14 | 24 | 0 | 0 | 0 | 0 | 38
    Part I: 45-64 years | 43 | 37 | 0 | 0 | 0 | 0 | 80
    Part I: 65 years and over | 18 | 22 | 0 | 0 | 0 | 0 | 40
    Part I: Not disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part II: number analyzed (Participants) | 0 | 0 | 38 | 1 | 13 | 6 | 58
    Part II: 18-44 years | 0 | 0 | 9 | 0 | 0 | 1 | 10
    Part II: 45-64 years | 0 | 0 | 19 | 0 | 7 | 4 | 30
    Part II: 65 years and over | 0 | 0 | 10 | 0 | 6 | 1 | 17
    Part II: Not disclosed | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sex/Gender, Customized [Count of Participants; unit: Participants] — Data for arm - Part II: Encorafenib + Binimetinib + Infigratinib is not disclosed to avoid risk of identification and kept under category Not disclosed category. Population: Number Analyzed for Part I and Part II = number of participants analyzed for reporting arms for respective parts. Part I and Part II participants are not exclusive.
  Participants
    Part I: number analyzed (Participants) | 75 | 83 | 0 | 0 | 0 | 0 | 158
    Part I: Female | 28 | 39 | 0 | 0 | 0 | 0 | 67
    Part I: Male | 47 | 44 | 0 | 0 | 0 | 0 | 91
    Part I: Not Disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part II: number analyzed (Participants) | 0 | 0 | 38 | 1 | 13 | 6 | 58
    Part II: Female | 0 | 0 | 22 | 0 | 5 | 1 | 28
    Part II: Male | 0 | 0 | 16 | 0 | 8 | 5 | 29
    Part II: Not Disclosed | 0 | 0 | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race is reported. Data for arm - Part II: Encorafenib + Binimetinib + Infigratinib is not disclosed to avoid risk of identification and kept under category Not disclosed category. Population: Number Analyzed for Part I and Part II = number of participants analyzed for reporting arms for respective parts. Part I and Part II participants are not exclusive.
  Participants
    Race: Part I: number analyzed (Participants) | 75 | 83 | 0 | 0 | 0 | 0 | 158
    Race: Part I: Caucasian | 74 | 82 | 0 | 0 | 0 | 0 | 156
    Race: Part I: Asian | 1 | 1 | 0 | 0 | 0 | 0 | 2
    Race: Part I: Not Disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Race: Part II: number analyzed (Participants) | 0 | 0 | 38 | 1 | 13 | 6 | 58
    Race: Part II: Caucasian | 0 | 0 | 37 | 0 | 13 | 6 | 56
    Race: Part II: Asian | 0 | 0 | 1 | 0 | 0 | 0 | 1
    Race: Part II: Not Disclosed | 0 | 0 | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity is reported. Data for arm - Part II: Encorafenib + Binimetinib + Infigratinib is not disclosed to avoid risk of identification and kept under category Not disclosed category. Population: Number Analyzed for Part I and Part II = number of participants analyzed for reporting arms for respective parts. Part I and Part II participants are not exclusive.
  Participants
    Ethnicity: Part I: number analyzed (Participants) | 75 | 83 | 0 | 0 | 0 | 0 | 158
    Ethnicity: Part I: Hispanic or Latino | 3 | 7 | 0 | 0 | 0 | 0 | 10
    Ethnicity: Part I: Not Hispanic or Latino | 72 | 76 | 0 | 0 | 0 | 0 | 148
    Ethnicity: Part I: Not Disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Ethnicity: Part II: number analyzed (Participants) | 0 | 0 | 38 | 1 | 13 | 6 | 58
    Ethnicity: Part II: Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 0 | 1
    Ethnicity: Part II: Not Hispanic or Latino | 0 | 0 | 37 | 0 | 13 | 6 | 56
    Ethnicity: Part II: Not Disclosed | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR): Part II
Description: ORR: percentage of participants with confirmed complete response (CR) and partial response (PR). Response evaluation criteria in solid tumors (RECIST) v1.1: a) CR = disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions that had a reduction in short axis to less than (<) 10 millimeter (mm). Disappearance of all non-target lesions. In addition, all lymph nodes assigned a non-target lesion must be non-pathological in size (<10 mm short axis) and b) PR = at least a 30 percent (%) decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. Any radiological assessments taken more than 30 days after the last dose of study therapy or after antineoplastic agents other than study treatments taken by the participants was excluded from the best overall response derivation. Confirmation of CR or PR was to be at least 4 weeks apart from the previous radiological assessment.
Time Frame: From the start of the treatment until disease/clinical progression or death or early study discontinuation, whichever happened earlier (maximum treatment exposure for Part II was 97.0 weeks)
Population: For Part II, full analysis set (FAS) consisted of all participants who received at least 1 dose of encorafenib or binimetinib or the assigned third agent following the assignment of the triple combination treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part II: Encorafenib + Binimetinib + Ribociclib | Part II: Encorafenib + Binimetinib + Infigratinib | Part II: Encorafenib + Binimetinib + Capmatinib | Part II: Encorafenib + Binimetinib + Buparlisib
Number analyzed (Participants) | 38 | 1 | 13 | 6
Percentage of participants | 2.6 [0.1 to 13.8] | 0 [NA to NA] — Only 1 participant evaluable. | 0 [0.0 to 24.7] | 0 [0.0 to 45.9]

2. Secondary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) in Cycle 1: Part II
Description: DLT was defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurred within the first cycle (first 21 days for infigratinib and capmatinib; 28 days for ribociclib and buparlisib) of treatment initiation and met the defined criteria for study.
Time Frame: Cycle 1 (21 days following the first dose of the combination treatment with buparlisib and capmatinib; 28 days for the combination with ribociclib and infigratinib)
Population: Dose-determining analysis set (DDS) consisted of all participants from the safety set for Part II who met the minimum requirements for safety evaluation and minimum exposure or experienced DLT during the first cycle of the assigned triple combination treatment. No participants were included in the dose-determining analysis set in the encorafenib/binimetinib+ infigratinib or buparlisib arm, hence no participants analyzed for these reporting arms for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Part II: Encorafenib + Binimetinib + Buparlisib: Participants, received encorafenib 450 mg (starting dose) once a day, binimetinib 45 mg (starting dose) twice a day and buparlisib 60 mg starting dose) once a day until disease progression or no clinical benefit. No dose reduction below 150 mg for encorafenib and 15 mg for binimetinib was permitted for this study. For buparlisib dose escalation was allowed till 100 mg and dose reduction was permitted till 30 mg. Treatment cycle for encorafenib, binimetinib and buparlisib was defined as 21 days of daily continuous treatment.
Arm/Group | Part II: Encorafenib + Binimetinib + Ribociclib | Part II: Encorafenib + Binimetinib + Infigratinib | Part II: Encorafenib + Binimetinib + Capmatinib | Part II: Encorafenib + Binimetinib + Buparlisib
Number analyzed (Participants) | 34 | 0 | 12 | 0
Participants | 1 |  | 0 |

3. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs): Part I
Description: An AE was defined as the appearance of (or worsening of any pre-existing) undesirable sign(s), symptom(s), or medical condition(s) that occurred after participants' signed informed consent has been obtained. An SAE was an AE resulting in any of the following outcomes: was fatal or life-threatening; resulted in persistent or significant disability/incapacity; constituted a congenital anomaly/birth defect; was medically significant; required inpatient hospitalization or prolongation of existing hospitalization. AEs included both SAEs and all Non-SAEs.
Time Frame: Day 1 up to 30 days after last dose (maximum treatment exposure for Part I was 403.7 weeks)
Population: Safety set included all participants who received at least 1 dose of encorafenib or binimetinib for Part I and had at least 1 valid post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Encorafenib + Binimetinib (Naive) | Part I: Encorafenib + Binimetinib (Non-naive)
Number analyzed (Participants) | 75 | 83
Participants
  AEs | 75 | 78
  SAEs | 47 | 37

4. Secondary Outcome: Number of Participants With AEs and SAEs: Part II
Description: as for outcome 3
Time Frame: Day 1 up to 30 days after last dose (maximum treatment exposure for Part II was 97.0 weeks)
Population: Safety set included all participants who received at least 1 dose of 3rd combination agent for Part II and had at least 1 valid post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part II: Encorafenib + Binimetinib + Ribociclib | Part II: Encorafenib + Binimetinib + Infigratinib | Part II: Encorafenib + Binimetinib + Capmatinib | Part II: Encorafenib + Binimetinib + Buparlisib
Number analyzed (Participants) | 38 | 1 | 13 | 6
Participants
  AEs | 37 | 1 | 12 | 6
  SAEs | 19 | 0 | 6 | 4

5. Secondary Outcome: Number of Participants With Worst Post-baseline Hematology Results Based on Common Terminology Criteria for Adverse Events (CTCAE) v4.03 Grade: Part I
Description: Parameters evaluated were: Activated partial thromboplastin time (APTT) (seconds [sec]) - CTCAE graded high, fibrinogen (gram per liter [g/L]) - CTCAE graded low, hemoglobin (g/L) - CTCAE graded low, hemoglobin (g/L) - CTCAE graded high, prothrombin international normalized ratio (PINR) - CTCAE graded high, lymphocytes (10^9 cells/L) - CTCAE graded low, lymphocytes (10^9 cells/L) - CTCAE graded high, neutrophils (10^9 cells/L) - CTCAE graded low, platelets (10^9 cells/L) - CTCAE graded low, leukocytes (10^9 cells/L) - CTCAE graded low, leukocytes (10^9 cells/L) - CTCAE graded high. CTCAE version 4.03 was used: grade 1 = mild, grade 2 = moderate, grade 3 = severe, grade 4 = life-threatening consequences; grade 0 = values not meeting any of the criteria for grade 1 or higher. Baseline = last non-missing value prior to the first dose of study treatment.
Time Frame: Baseline up to last dose (maximum treatment exposure for Part I was 403.7 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Encorafenib + Binimetinib (Naive) | Part I: Encorafenib + Binimetinib (Non-naive)
Number analyzed (Participants) | 75 | 83
Participants
  APTT -CTCAE graded high: Worst post-baseline value Grade 0 | 46 | 54
  APTT -CTCAE graded high: Worst post-baseline value Grade 1 | 1 | 4
  APTT -CTCAE graded high: Worst post-baseline value Grade 2 | 0 | 0
  APTT -CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 0
  APTT -CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0
  APTT -CTCAE graded high: Worst post-baseline value Missing | 28 | 25
  Fibrinogen - CTCAE graded low: Worst post-baseline value Grade 0 | 28 | 36
  Fibrinogen - CTCAE graded low: Worst post-baseline value Grade 1 | 8 | 9
  Fibrinogen - CTCAE graded low: Worst post-baseline value Grade 2 | 5 | 7
  Fibrinogen - CTCAE graded low: Worst post-baseline value Grade 3 | 4 | 1
  Fibrinogen - CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 0
  Fibrinogen - CTCAE graded low: Worst post-baseline value Missing | 30 | 30
  Hemoglobin - CTCAE graded low: Worst post-baseline value Grade 0 | 21 | 17
  Hemoglobin - CTCAE graded low: Worst post-baseline value Grade 1 | 28 | 39
  Hemoglobin - CTCAE graded low: Worst post-baseline value Grade 2 | 18 | 20
  Hemoglobin - CTCAE graded low: Worst post-baseline value Grade 3 | 8 | 6
  Hemoglobin - CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 0
  Hemoglobin - CTCAE graded low: Worst post-baseline value Missing | 0 | 1
  Hemoglobin - CTCAE graded high: Worst post-baseline value Grade 0 | 70 | 80
  Hemoglobin - CTCAE graded high: Worst post-baseline value Grade 1 | 4 | 2
  Hemoglobin - CTCAE graded high: Worst post-baseline value Grade 2 | 0 | 0
  Hemoglobin - CTCAE graded high: Worst post-baseline value Grade 3 | 1 | 0
  Hemoglobin - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0
  Hemoglobin - CTCAE graded high: Worst post-baseline value Missing | 0 | 1
  PINR -CTCAE graded high: Worst post-baseline value Grade 0 | 44 | 34
  PINR -CTCAE graded high: Worst post-baseline value Grade 1 | 0 | 2
  PINR -CTCAE graded high: Worst post-baseline value Grade 2 | 0 | 0
  PINR -CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 0
  PINR -CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0
  PINR -CTCAE graded high: Worst post-baseline value Missing | 31 | 47
  Lymphocytes - CTCAE graded low: Worst post-baseline value Grade 0 | 23 | 27
  Lymphocytes - CTCAE graded low: Worst post-baseline value Grade 1 | 22 | 24
  Lymphocytes - CTCAE graded low: Worst post-baseline value Grade 2 | 13 | 12
  Lymphocytes - CTCAE graded low: Worst post-baseline value Grade 3 | 6 | 10
  Lymphocytes - CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 1
  Lymphocytes - CTCAE graded low: Worst post-baseline value Missing | 11 | 9
  Lymphocytes - CTCAE graded high: Worst post-baseline value Grade 0 | 61 | 68
  Lymphocytes - CTCAE graded high: Worst post-baseline value Grade 1 | 0 | 0
  Lymphocytes - CTCAE graded high: Worst post-baseline value Grade 2 | 2 | 6
  Lymphocytes - CTCAE graded high: Worst post-baseline value Grade 3 | 1 | 0
  Lymphocytes - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0
  Lymphocytes - CTCAE graded high: Worst post-baseline value Missing | 11 | 9
  Neutrophils - CTCAE graded low: Worst post-baseline value Grade 0 | 52 | 62
  Neutrophils - CTCAE graded low: Worst post-baseline value Grade 1 | 4 | 6
  Neutrophils - CTCAE graded low: Worst post-baseline value Grade 2 | 5 | 4
  Neutrophils - CTCAE graded low: Worst post-baseline value Grade 3 | 3 | 1
  Neutrophils - CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 0
  Neutrophils - CTCAE graded low: Worst post-baseline value Missing | 11 | 10
  Platelets - CTCAE graded low: Worst post-baseline value Grade 0 | 59 | 71
  Platelets - CTCAE graded low: Worst post-baseline value Grade 1 | 14 | 11
  Platelets - CTCAE graded low: Worst post-baseline value Grade 2 | 2 | 0
  Platelets - CTCAE graded low: Worst post-baseline value Grade 3 | 0 | 0
  Platelets - CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 0
  Platelets - CTCAE graded low: Worst post-baseline value Missing | 0 | 1
  Leukocytes - CTCAE graded low: Worst post-baseline value Grade 0 | 52 | 61
  Leukocytes - CTCAE graded low: Worst post-baseline value Grade 1 | 11 | 14
  Leukocytes - CTCAE graded low: Worst post-baseline value Grade 2 | 3 | 3
  Leukocytes - CTCAE graded low: Worst post-baseline value Grade 3 | 0 | 0
  Leukocytes - CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 0
  Leukocytes - CTCAE graded low: Worst post-baseline value Missing | 9 | 5
  Leukocytes - CTCAE graded high: Worst post-baseline value Grade 0 | 66 | 78
  Leukocytes - CTCAE graded high: Worst post-baseline value Grade 1 | 0 | 0
  Leukocytes - CTCAE graded high: Worst post-baseline value Grade 2 | 0 | 0
  Leukocytes - CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 0
  Leukocytes - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0
  Leukocytes - CTCAE graded high: Worst post-baseline value Missing | 9 | 5

6. Secondary Outcome: Number of Participants With Worst Post-baseline Hematology Results Based on CTCAE v4.03 Grade: Part II
Description: Parameters evaluated were: APTT (sec) - CTCAE graded high, fibrinogen (g/L) - CTCAE graded low, hemoglobin (g/L) - CTCAE graded low, hemoglobin (g/L) - CTCAE graded high, PINR - CTCAE graded high, lymphocytes (10^9 cells/L) - CTCAE graded low, lymphocytes (10^9 cells/L) - CTCAE graded high, neutrophils (10^9 cells/L) - CTCAE graded low, platelets (10^9 cells/L) - CTCAE graded low, leukocytes (10^9 cells/L) - CTCAE graded low, leukocytes (10^9 cells/L) - CTCAE graded high. CTCAE version 4.03 was used: grade 1 = mild, grade 2 = moderate, grade 3 = severe, grade 4 = life-threatening consequences; grade 0 = values not meeting any of the criteria for grade 1 or higher. Baseline = last non-missing value prior to the first dose of study treatment in Part II.
Time Frame: Baseline up to last dose (maximum treatment exposure for Part II was 97.0 weeks)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part II: Encorafenib + Binimetinib + Ribociclib | Part II: Encorafenib + Binimetinib + Infigratinib | Part II: Encorafenib + Binimetinib + Capmatinib | Part II: Encorafenib + Binimetinib + Buparlisib
Number analyzed (Participants) | 38 | 1 | 13 | 6
Participants
  APTT- CTCAE graded high: Worst post-baseline value Grade 0 | 27 | 1 | 9 | 4
  APTT- CTCAE graded high: Worst post-baseline value Grade 1 | 0 | 0 | 0 | 0
  APTT- CTCAE graded high: Worst post-baseline value Grade 2 | 0 | 0 | 0 | 0
  APTT- CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 0 | 0 | 0
  APTT- CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  APTT- CTCAE graded high: Worst post-baseline value Missing | 11 | 0 | 4 | 2
  Fibrinogen: CTCAE graded low: Worst post-baseline value Grade 0 | 13 | 0 | 6 | 3
  Fibrinogen: CTCAE graded low: Worst post-baseline value Grade 1 | 3 | 1 | 1 | 0
  Fibrinogen: CTCAE graded low: Worst post-baseline value Grade 2 | 2 | 0 | 1 | 0
  Fibrinogen: CTCAE graded low: Worst post-baseline value Grade 3 | 1 | 0 | 0 | 0
  Fibrinogen: CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Fibrinogen: CTCAE graded low: Worst post-baseline value Missing | 19 | 0 | 5 | 3
  Hemoglobin- CTCAE graded low: Worst post-baseline value Grade 0 | 4 | 0 | 4 | 2
  Hemoglobin- CTCAE graded low: Worst post-baseline value Grade 1 | 15 | 1 | 5 | 1
  Hemoglobin- CTCAE graded low: Worst post-baseline value Grade 2 | 14 | 0 | 2 | 1
  Hemoglobin- CTCAE graded low: Worst post-baseline value Grade 3 | 4 | 0 | 1 | 2
  Hemoglobin- CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Hemoglobin- CTCAE graded low: Worst post-baseline value Missing | 1 | 0 | 1 | 0
  Hemoglobin- CTCAE graded high: Worst post-baseline value Grade 0 | 37 | 1 | 11 | 6
  Hemoglobin- CTCAE graded high: Worst post-baseline value Grade 1 | 0 | 0 | 1 | 0
  Hemoglobin- CTCAE graded high: Worst post-baseline value Grade 2 | 0 | 0 | 0 | 0
  Hemoglobin- CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 0 | 0 | 0
  Hemoglobin- CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Hemoglobin- CTCAE graded high: Worst post-baseline value Missing | 1 | 0 | 1 | 0
  PINR- CTCAE graded high: Worst post-baseline value Grade 0 | 14 | 1 | 8 | 1
  PINR- CTCAE graded high: Worst post-baseline value Grade 1 | 0 | 0 | 0 | 0
  PINR- CTCAE graded high: Worst post-baseline value Grade 2 | 0 | 0 | 0 | 0
  PINR- CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 0 | 0 | 0
  PINR- CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  PINR- CTCAE graded high: Worst post-baseline value Missing | 24 | 0 | 5 | 5
  Lymphocytes -CTCAE graded low: Worst post-baseline value Grade 0 | 5 | 0 | 4 | 2
  Lymphocytes -CTCAE graded low: Worst post-baseline value Grade 1 | 7 | 0 | 4 | 3
  Lymphocytes -CTCAE graded low: Worst post-baseline value Grade 2 | 9 | 0 | 3 | 1
  Lymphocytes -CTCAE graded low: Worst post-baseline value Grade 3 | 7 | 0 | 0 | 0
  Lymphocytes -CTCAE graded low: Worst post-baseline value Grade 4 | 1 | 0 | 0 | 0
  Lymphocytes -CTCAE graded low: Worst post-baseline value Missing | 9 | 1 | 2 | 0
  Lymphocytes- CTCAE graded high: Worst post-baseline value Grade 0 | 29 | 0 | 11 | 6
  Lymphocytes- CTCAE graded high: Worst post-baseline value Grade 1 | 0 | 0 | 0 | 0
  Lymphocytes- CTCAE graded high: Worst post-baseline value Grade 2 | 0 | 0 | 0 | 0
  Lymphocytes- CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 0 | 0 | 0
  Lymphocytes- CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Lymphocytes- CTCAE graded high: Worst post-baseline value Missing | 9 | 1 | 2 | 0
  Neutrophils- CTCAE graded low: Worst post-baseline value Grade 0 | 10 | 0 | 11 | 6
  Neutrophils- CTCAE graded low: Worst post-baseline value Grade 1 | 9 | 0 | 0 | 0
  Neutrophils- CTCAE graded low: Worst post-baseline value Grade 2 | 6 | 0 | 0 | 0
  Neutrophils- CTCAE graded low: Worst post-baseline value Grade 3 | 1 | 0 | 0 | 0
  Neutrophils- CTCAE graded low: Worst post-baseline value Grade 4 | 1 | 0 | 0 | 0
  Neutrophils- CTCAE graded low: Worst post-baseline value Missing | 11 | 1 | 2 | 0
  Platelets- CTCAE graded low: Worst post-baseline value Grade 0 | 33 | 1 | 11 | 6
  Platelets- CTCAE graded low: Worst post-baseline value Grade 1 | 4 | 0 | 1 | 0
  Platelets- CTCAE graded low: Worst post-baseline value Grade 2 | 0 | 0 | 0 | 0
  Platelets- CTCAE graded low: Worst post-baseline value Grade 3 | 0 | 0 | 0 | 0
  Platelets- CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Platelets- CTCAE graded low: Worst post-baseline value Missing | 1 | 0 | 1 | 0
  Leukocytes- CTCAE graded low: Worst post-baseline value Grade 0 | 8 | 0 | 11 | 6
  Leukocytes- CTCAE graded low: Worst post-baseline value Grade 1 | 8 | 0 | 0 | 0
  Leukocytes- CTCAE graded low: Worst post-baseline value Grade 2 | 12 | 0 | 0 | 0
  Leukocytes- CTCAE graded low: Worst post-baseline value Grade 3 | 3 | 0 | 0 | 0
  Leukocytes- CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Leukocytes- CTCAE graded low: Worst post-baseline value Missing | 7 | 1 | 2 | 0
  Leukocytes - CTCAE graded high: Worst post-baseline value Grade 0 | 31 | 0 | 11 | 6
  Leukocytes - CTCAE graded high: Worst post-baseline value Grade 1 | 0 | 0 | 0 | 0
  Leukocytes - CTCAE graded high: Worst post-baseline value Grade 2 | 0 | 0 | 0 | 0
  Leukocytes - CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 0 | 0 | 0
  Leukocytes - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Leukocytes - CTCAE graded high: Worst post-baseline value Missing | 7 | 1 | 2 | 0

7. Secondary Outcome: Number of Participants With Worst Post-baseline Serum Chemistry Results Based on CTCAE v4.03 Grade: Part I
Description: Parameters evaluated were: albumin (g/L)- CTCAE graded low, alkaline phosphatase (units per liter [U/L])- CTCAE graded high, alanine aminotransferase (U/L)- CTCAE graded high, amylase (U/L - CTCAE graded high, aspartate aminotransferase(U/L)- CTCAE graded high, bilirubin (micromole per liter [umol/L])- CTCAE graded high, creatinine (umol/L) - CTCAE graded high, creatine kinase (U/L)- CTCAE graded high, gamma glutamyl transferase (U/L)- CTCAE graded high, glucose (millimole per liter [mmol/L])- CTCAE graded low, high, potassium (mmol/L)- CTCAE graded low, potassium (mmol/L)- CTCAE graded high, magnesium (mmol/L)- CTCAE graded low, high, phosphate (mmol/L)- CTCAE graded low, sodium (mmol/L)- CTCAE graded low, sodium (mmol/L)- CTCAE graded high, urate (umol/L)- CTCAE graded high. CTCAE version 4.03 was used: grade 1 = mild, grade 2 = moderate, grade 3 = severe, grade 4 = life-threatening consequences; grade 0 = values not meeting any of the criteria for grade 1 or higher.
Time Frame: Baseline up to last dose (maximum treatment exposure for Part I was 403.7 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Encorafenib + Binimetinib (Naive) | Part I: Encorafenib + Binimetinib (Non-naive)
Number analyzed (Participants) | 75 | 83
Participants
  Albumin - CTCAE graded low: Worst post-baseline value Grade 0 | 32 | 40
  Albumin - CTCAE graded low: Worst post-baseline value Grade 1 | 35 | 29
  Albumin - CTCAE graded low: Worst post-baseline value Grade 2 | 8 | 12
  Albumin - CTCAE graded low: Worst post-baseline value Grade 3 | 0 | 1
  Albumin - CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 0
  Albumin - CTCAE graded low: Worst post-baseline value Missing | 0 | 1
  Alkaline Phosphatase - CTCAE graded high: Worst post-baseline value Grade 0 | 39 | 43
  Alkaline Phosphatase - CTCAE graded high: Worst post-baseline value Grade 1 | 28 | 31
  Alkaline Phosphatase - CTCAE graded high: Worst post-baseline value Grade 2 | 5 | 5
  Alkaline Phosphatase - CTCAE graded high: Worst post-baseline value Grade 3 | 3 | 3
  Alkaline Phosphatase - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0
  Alkaline Phosphatase - CTCAE graded high: Worst post-baseline value Missing | 0 | 1
  Alanine Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 0 | 38 | 51
  Alanine Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 1 | 27 | 28
  Alanine Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 2 | 5 | 2
  Alanine Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 3 | 5 | 0
  Alanine Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0
  Alanine Aminotransferase - CTCAE graded high: Worst post-baseline value Missing | 0 | 2
  Amylase - CTCAE graded high: Worst post-baseline value Grade 0 | 53 | 52
  Amylase - CTCAE graded high: Worst post-baseline value Grade 1 | 14 | 6
  Amylase - CTCAE graded high: Worst post-baseline value Grade 2 | 5 | 2
  Amylase - CTCAE graded high: Worst post-baseline value Grade 3 | 2 | 2
  Amylase - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 1
  Amylase - CTCAE graded high: Worst post-baseline value Missing | 1 | 20
  Aspartate Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 0 | 38 | 50
  Aspartate Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 1 | 30 | 29
  Aspartate Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 2 | 4 | 2
  Aspartate Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 3 | 3 | 1
  Aspartate Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0
  Aspartate Aminotransferase - CTCAE graded high: Worst post-baseline value Missing | 0 | 1
  Bilirubin - CTCAE graded high: Worst post-baseline value Grade 0 | 73 | 81
  Bilirubin - CTCAE graded high: Worst post-baseline value Grade 1 | 1 | 0
  Bilirubin - CTCAE graded high: Worst post-baseline value Grade 2 | 1 | 0
  Bilirubin - CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 1
  Bilirubin - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0
  Bilirubin - CTCAE graded high: Worst post-baseline value Missing | 0 | 1
  Creatine Kinase - CTCAE graded high: Worst post-baseline value Grade 0 | 22 | 56
  Creatine Kinase - CTCAE graded high: Worst post-baseline value Grade 1 | 30 | 15
  Creatine Kinase - CTCAE graded high: Worst post-baseline value Grade 2 | 18 | 8
  Creatine Kinase - CTCAE graded high: Worst post-baseline value Grade 3 | 4 | 2
  Creatine Kinase - CTCAE graded high: Worst post-baseline value Grade 4 | 1 | 1
  Creatine Kinase - CTCAE graded high: Worst post-baseline value Missing | 0 | 1
  Creatinine - CTCAE graded high: Worst post-baseline value Grade 0 | 2 | 4
  Creatinine - CTCAE graded high: Worst post-baseline value Grade 1 | 57 | 56
  Creatinine - CTCAE graded high: Worst post-baseline value Grade 2 | 14 | 22
  Creatinine - CTCAE graded high: Worst post-baseline value Grade 3 | 2 | 0
  Creatinine - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0
  Creatinine - CTCAE graded high: Worst post-baseline value Missing | 0 | 1
  Gamma Glutamyl Transferase - CTCAE graded high: Worst post-baseline value Grade 0 | 20 | 33
  Gamma Glutamyl Transferase - CTCAE graded high: Worst post-baseline value Grade 1 | 19 | 18
  Gamma Glutamyl Transferase - CTCAE graded high: Worst post-baseline value Grade 2 | 14 | 13
  Gamma Glutamyl Transferase - CTCAE graded high: Worst post-baseline value Grade 3 | 20 | 15
  Gamma Glutamyl Transferase - CTCAE graded high: Worst post-baseline value Grade 4 | 2 | 3
  Gamma Glutamyl Transferase - CTCAE graded high: Worst post-baseline value Missing | 0 | 1
  Glucose - CTCAE graded low: Worst post-baseline value Grade 0 | 55 | 67
  Glucose - CTCAE graded low: Worst post-baseline value Grade 1 | 15 | 7
  Glucose - CTCAE graded low: Worst post-baseline value Grade 2 | 1 | 1
  Glucose - CTCAE graded low: Worst post-baseline value Grade 3 | 0 | 0
  Glucose - CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 0
  Glucose - CTCAE graded low: Worst post-baseline value Missing | 4 | 8
  Glucose - CTCAE graded high: Worst post-baseline value Grade 0 | 56 | 60
  Glucose - CTCAE graded high: Worst post-baseline value Grade 1 | 4 | 10
  Glucose - CTCAE graded high: Worst post-baseline value Grade 2 | 3 | 0
  Glucose - CTCAE graded high: Worst post-baseline value Grade 3 | 7 | 5
  Glucose - CTCAE graded high: Worst post-baseline value Grade 4 | 1 | 0
  Glucose - CTCAE graded high: Worst post-baseline value Missing | 4 | 8
  Potassium - CTCAE graded low: Worst post-baseline value Grade 0 | 65 | 74
  Potassium - CTCAE graded low: Worst post-baseline value Grade 1 | 7 | 5
  Potassium - CTCAE graded low: Worst post-baseline value Grade 2 | 0 | 0
  Potassium - CTCAE graded low: Worst post-baseline value Grade 3 | 3 | 3
  Potassium - CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 0
  Potassium - CTCAE graded low: Worst post-baseline value Missing | 0 | 1
  Potassium - CTCAE graded high: Worst post-baseline value Grade 0 | 54 | 66
  Potassium - CTCAE graded high: Worst post-baseline value Grade 1 | 18 | 15
  Potassium - CTCAE graded high: Worst post-baseline value Grade 2 | 2 | 0
  Potassium - CTCAE graded high: Worst post-baseline value Grade 3 | 1 | 0
  Potassium - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 1
  Potassium - CTCAE graded high: Worst post-baseline value Missing | 0 | 1
  Magnesium - CTCAE graded low: Worst post-baseline value Grade 0 | 66 | 68
  Magnesium - CTCAE graded low: Worst post-baseline value Grade 1 | 8 | 14
  Magnesium - CTCAE graded low: Worst post-baseline value Grade 2 | 0 | 0
  Magnesium - CTCAE graded low: Worst post-baseline value Grade 3 | 1 | 0
  Magnesium - CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 0
  Magnesium - CTCAE graded low: Worst post-baseline value Missing | 0 | 1
  Magnesium - CTCAE graded high: Worst post-baseline value Grade 0 | 74 | 79
  Magnesium - CTCAE graded high: Worst post-baseline value Grade 1 | 1 | 3
  Magnesium - CTCAE graded high: Worst post-baseline value Grade 2 | 0 | 0
  Magnesium - CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 0
  Magnesium - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0
  Magnesium - CTCAE graded high: Worst post-baseline value Missing | 0 | 1
  Phosphate - CTCAE graded low: Worst post-baseline value Grade 0 | 40 | 62
  Phosphate - CTCAE graded low: Worst post-baseline value Grade 1 | 3 | 3
  Phosphate - CTCAE graded low: Worst post-baseline value Grade 2 | 24 | 12
  Phosphate - CTCAE graded low: Worst post-baseline value Grade 3 | 8 | 4
  Phosphate - CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 1
  Phosphate - CTCAE graded low: Worst post-baseline value Missing | 0 | 1
  Sodium - CTCAE graded low: Worst post-baseline value Grade 0 | 54 | 53
  Sodium - CTCAE graded low: Worst post-baseline value Grade 1 | 21 | 24
  Sodium - CTCAE graded low: Worst post-baseline value Grade 2 | 0 | 0
  Sodium - CTCAE graded low: Worst post-baseline value Grade 3 | 0 | 5
  Sodium - CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 0
  Sodium - CTCAE graded low: Worst post-baseline value Missing | 0 | 1
  Sodium - CTCAE graded high: Worst post-baseline value Grade 0 | 66 | 75
  Sodium - CTCAE graded high: Worst post-baseline value Grade 1 | 9 | 6
  Sodium - CTCAE graded high: Worst post-baseline value Grade 2 | 0 | 1
  Sodium - CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 0
  Sodium - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0
  Sodium - CTCAE graded high: Worst post-baseline value Missing | 0 | 1
  Urate - CTCAE graded high: Worst post-baseline value Grade 0 | 75 | 82
  Urate - CTCAE graded high: Worst post-baseline value Grade 1 | 0 | 0
  Urate - CTCAE graded high: Worst post-baseline value Grade 2 | 0 | 0
  Urate - CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 0
  Urate - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0
  Urate - CTCAE graded high: Worst post-baseline value Missing | 0 | 1

8. Secondary Outcome: Number of Participants With Worst Post-baseline Serum Chemistry Results Based on CTCAE v4.03 Grade: Part II
Description: Parameters evaluated were: albumin (g/L)- CTCAE graded low, alkaline phosphatase (U/L)- CTCAE graded high, alanine aminotransferase (U/L)- CTCAE graded high, amylase (U/L) - CTCAE graded high, aspartate aminotransferase(U/L)- CTCAE graded high, bilirubin (umol/L)- CTCAE graded high, creatinine (umol/L) - CTCAE graded high, creatine kinase (U/L)- CTCAE graded high, gamma glutamyl transferase (U/L)- CTCAE graded high, glucose (mmol/L)- CTCAE graded low, high, potassium (mmol/L)- CTCAE graded low, potassium (mmol/L)- CTCAE graded high, magnesium (mmol/L)- CTCAE graded low, high, phosphate (mmol/L)- CTCAE graded low, sodium (mmol/L)- CTCAE graded low, sodium (mmol/L)- CTCAE graded high, urate (umol/L)- CTCAE graded high. CTCAE version 4.03 was used: grade 1 = mild, grade 2 = moderate, grade 3 = severe, grade 4 = life-threatening consequences; grade 0 = values not meeting any of the criteria for grade 1 or higher.
Time Frame: Baseline up to last dose (maximum treatment exposure for Part II was 97.0 weeks)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part II: Encorafenib + Binimetinib + Ribociclib | Part II: Encorafenib + Binimetinib + Infigratinib | Part II: Encorafenib + Binimetinib + Capmatinib | Part II: Encorafenib + Binimetinib + Buparlisib
Number analyzed (Participants) | 38 | 1 | 13 | 6
Participants
  Albumin- CTCAE graded low: Worst post-baseline value Grade 0 | 16 | 1 | 1 | 3
  Albumin- CTCAE graded low: Worst post-baseline value Grade 1 | 13 | 0 | 6 | 0
  Albumin- CTCAE graded low: Worst post-baseline value Grade 2 | 7 | 0 | 3 | 1
  Albumin- CTCAE graded low: Worst post-baseline value Grade 3 | 1 | 0 | 2 | 1
  Albumin- CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Albumin- CTCAE graded low: Worst post-baseline value Missing | 1 | 0 | 1 | 1
  Alkaline Phosphatase - CTCAE graded high: Worst post-baseline value Grade 0 | 22 | 1 | 7 | 1
  Alkaline Phosphatase - CTCAE graded high: Worst post-baseline value Grade 1 | 10 | 0 | 3 | 4
  Alkaline Phosphatase - CTCAE graded high: Worst post-baseline value Grade 2 | 3 | 0 | 2 | 1
  Alkaline Phosphatase - CTCAE graded high: Worst post-baseline value Grade 3 | 2 | 0 | 0 | 0
  Alkaline Phosphatase - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Alkaline Phosphatase - CTCAE graded high: Worst post-baseline value Missing | 1 | 0 | 1 | 0
  Alanine Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 0 | 27 | 1 | 9 | 4
  Alanine Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 1 | 6 | 0 | 2 | 1
  Alanine Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 2 | 2 | 0 | 0 | 0
  Alanine Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 3 | 1 | 0 | 1 | 0
  Alanine Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 4 | 1 | 0 | 0 | 1
  Alanine Aminotransferase - CTCAE graded high: Worst post-baseline value Missing | 1 | 0 | 1 | 0
  Amylase - CTCAE graded high: Worst post-baseline value Grade 0 | 27 | 1 | 9 | 1
  Amylase - CTCAE graded high: Worst post-baseline value Grade 1 | 1 | 0 | 2 | 0
  Amylase - CTCAE graded high: Worst post-baseline value Grade 2 | 0 | 0 | 0 | 1
  Amylase - CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 0 | 0 | 0
  Amylase - CTCAE graded high: Worst post-baseline value Grade 4 | 2 | 0 | 0 | 0
  Amylase - CTCAE graded high: Worst post-baseline value Missing | 8 | 0 | 2 | 4
  Aspartate Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 0 | 27 | 1 | 8 | 3
  Aspartate Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 1 | 6 | 0 | 4 | 2
  Aspartate Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 2 | 3 | 0 | 0 | 0
  Aspartate Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 3 | 1 | 0 | 0 | 1
  Aspartate Aminotransferase - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase - CTCAE graded high: Worst post-baseline value Missing | 1 | 0 | 1 | 0
  Bilirubin - CTCAE graded high: Worst post-baseline value Grade 0 | 37 | 1 | 12 | 6
  Bilirubin - CTCAE graded high: Worst post-baseline value Grade 1 | 0 | 0 | 0 | 0
  Bilirubin - CTCAE graded high: Worst post-baseline value Grade 2 | 0 | 0 | 0 | 0
  Bilirubin - CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 0 | 0 | 0
  Bilirubin - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Bilirubin - CTCAE graded high: Worst post-baseline value Missing | 1 | 0 | 1 | 0
  Creatine Kinase - CTCAE graded high: Worst post-baseline value Grade 0 | 20 | 0 | 6 | 3
  Creatine Kinase - CTCAE graded high: Worst post-baseline value Grade 1 | 14 | 1 | 4 | 2
  Creatine Kinase - CTCAE graded high: Worst post-baseline value Grade 2 | 3 | 0 | 0 | 0
  Creatine Kinase - CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 0 | 2 | 0
  Creatine Kinase - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Creatine Kinase - CTCAE graded high: Worst post-baseline value Missing | 1 | 0 | 1 | 1
  Creatinine - CTCAE graded high: Worst post-baseline value Grade 0 | 1 | 0 | 0 | 1
  Creatinine - CTCAE graded high: Worst post-baseline value Grade 1 | 25 | 1 | 4 | 3
  Creatinine - CTCAE graded high: Worst post-baseline value Grade 2 | 11 | 0 | 8 | 1
  Creatinine - CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 0 | 0 | 0
  Creatinine - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Creatinine - CTCAE graded high: Worst post-baseline value Missing | 1 | 0 | 1 | 1
  Gamma Glutamyl Transferase - CTCAE graded high: Worst post-baseline value Grade 0 | 20 | 1 | 5 | 0
  Gamma Glutamyl Transferase - CTCAE graded high: Worst post-baseline value Grade 1 | 9 | 0 | 2 | 1
  Gamma Glutamyl Transferase - CTCAE graded high: Worst post-baseline value Grade 2 | 1 | 0 | 2 | 2
  Gamma Glutamyl Transferase - CTCAE graded high: Worst post-baseline value Grade 3 | 7 | 0 | 3 | 3
  Gamma Glutamyl Transferase - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Gamma Glutamyl Transferase - CTCAE graded high: Worst post-baseline value Missing | 1 | 0 | 1 | 0
  Glucose - CTCAE graded low: Worst post-baseline value Grade 0 | 24 | 0 | 11 | 5
  Glucose - CTCAE graded low: Worst post-baseline value Grade 1 | 6 | 1 | 1 | 0
  Glucose - CTCAE graded low: Worst post-baseline value Grade 2 | 0 | 0 | 0 | 0
  Glucose - CTCAE graded low: Worst post-baseline value Grade 3 | 0 | 0 | 0 | 0
  Glucose - CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Glucose - CTCAE graded low: Worst post-baseline value Missing | 8 | 0 | 1 | 1
  Glucose - CTCAE graded high: Worst post-baseline value Grade 0 | 26 | 1 | 10 | 4
  Glucose - CTCAE graded high: Worst post-baseline value Grade 1 | 2 | 0 | 1 | 1
  Glucose - CTCAE graded high: Worst post-baseline value Grade 2 | 0 | 0 | 0 | 0
  Glucose - CTCAE graded high: Worst post-baseline value Grade 3 | 1 | 0 | 1 | 0
  Glucose - CTCAE graded high: Worst post-baseline value Grade 4 | 1 | 0 | 0 | 0
  Glucose - CTCAE graded high: Worst post-baseline value Missing | 8 | 0 | 1 | 1
  Potassium - CTCAE graded low: Worst post-baseline value Grade 0 | 34 | 1 | 11 | 5
  Potassium - CTCAE graded low: Worst post-baseline value Grade 1 | 3 | 0 | 1 | 0
  Potassium - CTCAE graded low: Worst post-baseline value Grade 2 | 0 | 0 | 0 | 0
  Potassium - CTCAE graded low: Worst post-baseline value Grade 3 | 0 | 0 | 0 | 0
  Potassium - CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Potassium - CTCAE graded low: Worst post-baseline value Missing | 1 | 0 | 1 | 1
  Potassium - CTCAE graded high: Worst post-baseline value Grade 0 | 32 | 1 | 9 | 3
  Potassium - CTCAE graded high: Worst post-baseline value Grade 1 | 4 | 0 | 3 | 2
  Potassium - CTCAE graded high: Worst post-baseline value Grade 2 | 1 | 0 | 0 | 0
  Potassium - CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 0 | 0 | 0
  Potassium - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Potassium - CTCAE graded high: Worst post-baseline value Missing | 1 | 0 | 1 | 1
  Magnesium - CTCAE graded low: Worst post-baseline value Grade 0 | 35 | 1 | 10 | 4
  Magnesium - CTCAE graded low: Worst post-baseline value Grade 1 | 2 | 0 | 2 | 1
  Magnesium - CTCAE graded low: Worst post-baseline value Grade 2 | 0 | 0 | 0 | 0
  Magnesium - CTCAE graded low: Worst post-baseline value Grade 3 | 0 | 0 | 0 | 0
  Magnesium - CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Magnesium - CTCAE graded low: Worst post-baseline value Missing | 1 | 0 | 1 | 1
  Magnesium - CTCAE graded high: Worst post-baseline value Grade 0 | 36 | 1 | 12 | 5
  Magnesium - CTCAE graded high: Worst post-baseline value Grade 1 | 1 | 0 | 0 | 0
  Magnesium - CTCAE graded high: Worst post-baseline value Grade 2 | 0 | 0 | 0 | 0
  Magnesium - CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 0 | 0 | 0
  Magnesium - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Magnesium - CTCAE graded high: Worst post-baseline value Missing | 1 | 0 | 1 | 1
  Phosphate - CTCAE graded low: Worst post-baseline value Grade 0 | 25 | 1 | 7 | 4
  Phosphate - CTCAE graded low: Worst post-baseline value Grade 1 | 2 | 0 | 1 | 1
  Phosphate - CTCAE graded low: Worst post-baseline value Grade 2 | 7 | 0 | 3 | 0
  Phosphate - CTCAE graded low: Worst post-baseline value Grade 3 | 1 | 0 | 1 | 0
  Phosphate - CTCAE graded low: Worst post-baseline value Grade 4 | 2 | 0 | 0 | 0
  Phosphate - CTCAE graded low: Worst post-baseline value Missing | 1 | 0 | 1 | 1
  Sodium -CTCAE graded low: Worst post-baseline value Grade 0 | 28 | 1 | 10 | 3
  Sodium -CTCAE graded low: Worst post-baseline value Grade 1 | 7 | 0 | 2 | 2
  Sodium -CTCAE graded low: Worst post-baseline value Grade 2 | 0 | 0 | 0 | 0
  Sodium -CTCAE graded low: Worst post-baseline value Grade 3 | 2 | 0 | 0 | 0
  Sodium -CTCAE graded low: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Sodium -CTCAE graded low: Worst post-baseline value Missing | 1 | 0 | 1 | 1
  Sodium - CTCAE graded high: Worst post-baseline value Grade 0 | 35 | 1 | 12 | 4
  Sodium - CTCAE graded high: Worst post-baseline value Grade 1 | 2 | 0 | 0 | 1
  Sodium - CTCAE graded high: Worst post-baseline value Grade 2 | 0 | 0 | 0 | 0
  Sodium - CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 0 | 0 | 0
  Sodium - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Sodium - CTCAE graded high: Worst post-baseline value Missing | 1 | 0 | 1 | 1
  Urate - CTCAE graded high: Worst post-baseline value Grade 0 | 37 | 1 | 12 | 5
  Urate - CTCAE graded high: Worst post-baseline value Grade 1 | 0 | 0 | 0 | 0
  Urate - CTCAE graded high: Worst post-baseline value Grade 2 | 0 | 0 | 0 | 0
  Urate - CTCAE graded high: Worst post-baseline value Grade 3 | 0 | 0 | 0 | 0
  Urate - CTCAE graded high: Worst post-baseline value Grade 4 | 0 | 0 | 0 | 0
  Urate - CTCAE graded high: Worst post-baseline value Missing | 1 | 0 | 1 | 1

9. Secondary Outcome: Number of Participants With Newly Occurring Notably Abnormal Vital Signs: Part I
Description: Vital signs evaluated were: Low/high systolic blood pressure (BP) (millimeter of Mercury [mmHg]): less than or equal to (<=) 90 mmHg with decrease from baseline of >=20 mmHg / >=160 mmHg with increase from baseline of >=20 mmHg; low/high diastolic BP [mmHg]: <=50 mmHg with decrease from baseline of >=15 mmHg / >=100 mmHg with increase from baseline of >=15 mmHg; low/high pulse rate (beats per minute [bpm]): <=50 bpm with decrease from baseline of >=15 bpm / >=120 bpm with increase from baseline of >=15 bpm; low/high weight (kilogram [kg]): >=20% decrease/increase from baseline; and low/high body temperature (degree Celsius [C]): <=36 C / >= 37.5 C.
Time Frame: During study treatment (maximum treatment exposure for Part I was 403.7 weeks)
Population: Safety set included all participants who received at least 1 dose of encorafenib or binimetinib for Part I and had at least 1 valid post-baseline safety assessment. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Encorafenib + Binimetinib (Naive) | Part I: Encorafenib + Binimetinib (Non-naive)
Number analyzed (Participants) | 75 | 83
Participants
  Sitting Pulse Rate: High: number analyzed (Participants) | 75 | 79
  Sitting Pulse Rate: High | 2 | 8
  Sitting Pulse Rate: Low: number analyzed (Participants) | 75 | 80
  Sitting Pulse Rate: Low | 5 | 4
  Sitting Systolic BP: High: number analyzed (Participants) | 74 | 80
  Sitting Systolic BP: High | 18 | 5
  Sitting Systolic BP: Low: number analyzed (Participants) | 75 | 78
  Sitting Systolic BP: Low | 3 | 2
  Sitting Diastolic BP: High: number analyzed (Participants) | 75 | 79
  Sitting Diastolic BP: High | 11 | 4
  Sitting Diastolic BP: Low: number analyzed (Participants) | 74 | 80
  Sitting Diastolic BP: Low | 5 | 3
  Weight: High: number analyzed (Participants) | 74 | 71
  Weight: High | 0 | 2
  Weight: Low: number analyzed (Participants) | 74 | 71
  Weight: Low | 0 | 0
  Body temperature: High: number analyzed (Participants) | 74 | 79
  Body temperature: High | 14 | 14
  Body temperature: Low: number analyzed (Participants) | 60 | 71
  Body temperature: Low | 44 | 36

10. Secondary Outcome: Number of Participants With Newly Occurring Notably Abnormal Vital Signs: Part II
Description: Vital signs evaluated were: Low/high systolic BP (mmHg): <=90 mmHg with decrease from baseline of >=20 mmHg / >=160 mmHg with increase from baseline of >=20 mmHg; low/high diastolic BP [mmHg]: <=50 mmHg with decrease from baseline of >=15 mmHg / >=100 mmHg with increase from baseline of >=15 mmHg; low/high pulse rate (bpm): <=50 bpm with decrease from baseline of >=15 bpm / >=120 bpm with increase from baseline of >=15 bpm; low/high weight (kg): >=20% decrease/increase from baseline; and low/high body temperature (C): <=36 C / >= 37.5 C.
Time Frame: During study treatment (maximum treatment exposure for Part II was 97.0 weeks)
Population: Safety set included all participants who received at least 1 dose of 3rd combination agent for Part II and had at least 1 valid post-baseline safety assessment. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Part II: Encorafenib + Binimetinib + Ribociclib | Part II: Encorafenib + Binimetinib + Infigratinib | Part II: Encorafenib + Binimetinib + Capmatinib | Part II: Encorafenib + Binimetinib + Buparlisib
Number analyzed (Participants) | 38 | 1 | 13 | 6
Participants
  Sitting Pulse Rate: High: number analyzed (Participants) | 37 | 1 | 13 | 6
  Sitting Pulse Rate: High | 2 | 0 | 0 | 1
  Sitting Pulse Rate: Low: number analyzed (Participants) | 37 | 1 | 13 | 6
  Sitting Pulse Rate: Low | 1 | 0 | 0 | 0
  Sitting Systolic BP: High: number analyzed (Participants) | 37 | 1 | 11 | 6
  Sitting Systolic BP: High | 2 | 0 | 4 | 0
  Sitting Systolic BP: Low: number analyzed (Participants) | 37 | 1 | 13 | 6
  Sitting Systolic BP: Low | 0 | 0 | 0 | 0
  Sitting Diastolic BP: High: number analyzed (Participants) | 37 | 1 | 13 | 6
  Sitting Diastolic BP: High | 2 | 0 | 1 | 0
  Sitting Diastolic BP: Low: number analyzed (Participants) | 37 | 1 | 13 | 6
  Sitting Diastolic BP: Low | 1 | 0 | 0 | 0
  Weight: High: number analyzed (Participants) | 36 | 1 | 13 | 5
  Weight: High | 0 | 0 | 0 | 0
  Weight: Low: number analyzed (Participants) | 36 | 1 | 13 | 5
  Weight: Low | 1 | 0 | 0 | 0
  Body temperature: High: number analyzed (Participants) | 36 | 1 | 13 | 6
  Body temperature: High | 3 | 0 | 1 | 1
  Body temperature: Low: number analyzed (Participants) | 30 | 1 | 11 | 5
  Body temperature: Low | 14 | 1 | 6 | 3

11. Secondary Outcome: Number of Participants With Notable Electrocardiograms (ECG) Values: Part I
Description: Number of participants with notable ECG values were reported in this outcome measure. Abnormality categories were: Heart rate (HR): increase from baseline >25% and to a value >100 bpm, decrease from baseline >25% and to a value <60 bpm; PR: increase from baseline >25% and to a value >200 millisecond (ms); QRS: increase from baseline >25% and to a value >110 ms; QT: increase from baseline >30 ms, increase from baseline >60 ms, new interval >450 ms, new interval >480 ms, new interval >500 ms; and Corrected QT interval by Fridericia (QTcF): increase from baseline >30 ms, increase from baseline >60 ms, new interval >450 ms, new interval >480 ms, new interval >500 ms. New = newly occurred post-baseline value.
Time Frame: During study treatment (maximum treatment exposure for Part I was 403.7 weeks)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Encorafenib + Binimetinib (Naive) | Part I: Encorafenib + Binimetinib (Non-naive)
Number analyzed (Participants) | 75 | 83
Participants
  HR: Increase from baseline >25% & to a value >100 bpm: number analyzed (Participants) | 74 | 80
  HR: Increase from baseline >25% & to a value >100 bpm | 10 | 5
  HR: Decrease from baseline >25% & to a value <60 bpm: number analyzed (Participants) | 74 | 80
  HR: Decrease from baseline >25% & to a value <60 bpm | 37 | 23
  PR: Increase from baseline >25% & to a value >200 ms: number analyzed (Participants) | 72 | 80
  PR: Increase from baseline >25% & to a value >200 ms | 5 | 1
  QRS: Increase from baseline >25% & to a value >110 ms: number analyzed (Participants) | 75 | 80
  QRS: Increase from baseline >25% & to a value >110 ms | 3 | 0
  QT: Increase from baseline >30 ms: number analyzed (Participants) | 75 | 80
  QT: Increase from baseline >30 ms | 61 | 48
  QT: Increase from baseline >60 ms: number analyzed (Participants) | 75 | 80
  QT: Increase from baseline >60 ms | 29 | 15
  QT: New Interval >450 ms: number analyzed (Participants) | 75 | 78
  QT: New Interval >450 ms | 24 | 4
  QT: New Interval >480 ms: number analyzed (Participants) | 75 | 80
  QT: New Interval >480 ms | 5 | 3
  QT: New Interval >500 ms: number analyzed (Participants) | 75 | 80
  QT: New Interval >500 ms | 3 | 0
  QTcF: Increase from baseline >30 ms: number analyzed (Participants) | 75 | 80
  QTcF: Increase from baseline >30 ms | 46 | 31
  QTcF: Increase from baseline >60 ms: number analyzed (Participants) | 75 | 80
  QTcF: Increase from baseline >60 ms | 4 | 2
  QTcF: New Interval >450 ms: number analyzed (Participants) | 74 | 77
  QTcF: New Interval >450 ms | 28 | 15
  QTcF: New Interval >480 ms: number analyzed (Participants) | 75 | 80
  QTcF: New Interval >480 ms | 4 | 0
  QTcF: New Interval >500 ms: number analyzed (Participants) | 75 | 80
  QTcF: New Interval >500 ms | 1 | 0

12. Secondary Outcome: Number of Participants With Notable ECG Values: Part II
Description: Number of participants with notable ECG values were reported in this outcome measure. Abnormality categories were: HR: increase from baseline >25% and to a value >100 bpm, decrease from baseline >25% and to a value <60 bpm; PR: increase from baseline >25% and to a value >200 ms; QRS: increase from baseline >25% and to a value >110 ms; QT: increase from baseline >30 ms, increase from baseline >60 ms, new interval >450 ms, new interval >480 ms, new interval >500 ms; and QTcF: increase from baseline >30 ms, increase from baseline >60 ms, new interval >450 ms, new interval >480 ms, new interval >500 ms. New = newly occurred post-baseline value.
Time Frame: During study treatment (maximum treatment exposure for Part II was 97.0 weeks)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part II: Encorafenib + Binimetinib + Ribociclib | Part II: Encorafenib + Binimetinib + Infigratinib | Part II: Encorafenib + Binimetinib + Capmatinib | Part II: Encorafenib + Binimetinib + Buparlisib
Number analyzed (Participants) | 38 | 1 | 13 | 6
Participants
  HR: Increase from baseline >25% & to a value >100 bpm | 3 | 0 | 2 | 1
  HR: Decrease from baseline >25% & to a value <60 bpm | 14 | 0 | 7 | 0
  PR: Increase from baseline >25% & to a value >200 ms: number analyzed (Participants) | 37 | 1 | 13 | 6
  PR: Increase from baseline >25% & to a value >200 ms | 1 | 0 | 2 | 0
  QRS: Increase from baseline >25% & to a value >110 ms | 0 | 0 | 0 | 0
  QT: Increase from baseline >30 ms | 24 | 0 | 9 | 0
  QT: Increase from baseline >60 ms | 2 | 0 | 0 | 0
  QT: New Interval >450 ms: number analyzed (Participants) | 37 | 0 | 13 | 6
  QT: New Interval >450 ms | 3 |  | 3 | 0
  QT: New Interval >480 ms | 1 | 0 | 0 | 0
  QT: New Interval >500 ms | 0 | 0 | 0 | 0
  QTcF: Increase from baseline >30 ms | 11 | 0 | 2 | 1
  QTcF: Increase from baseline >60 ms | 0 | 0 | 0 | 0
  QTcF: New Interval >450 ms: number analyzed (Participants) | 37 | 1 | 13 | 5
  QTcF: New Interval >450 ms | 14 | 0 | 3 | 0
  QTcF: New Interval >480 ms | 0 | 0 | 0 | 0
  QTcF: New Interval >500 ms | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With At Least One Dose Interruption: Part I
Description: In this outcome measure number of participants with at least 1 dose interruption for encorafenib and binimetinib were reported.
Time Frame: During study treatment (maximum treatment exposure for Part I was 403.7 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Encorafenib + Binimetinib (Naive) | Part I: Encorafenib + Binimetinib (Non-naive)
Number analyzed (Participants) | 75 | 83
Participants
  Encorafenib | 46 | 40
  Binimetinib | 44 | 41

14. Secondary Outcome: Number of Participants With At Least One Dose Interruption: Part II
Description: In this outcome measure number of participants with at least 1 dose interruption for encorafenib, binimetinib, and each third combination agent were reported.
Time Frame: During study treatment (maximum treatment exposure for Part II was 97.0 weeks)
Population: Safety set included all participants who received at least 1 dose of 3rd combination agent for Part II and had at least 1 valid post-baseline safety assessment. Here, "Number Analyzed" signifies number of participants evaluable for specified treatment in the respective reporting arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Part II: Encorafenib + Binimetinib + Ribociclib | Part II: Encorafenib + Binimetinib + Infigratinib | Part II: Encorafenib + Binimetinib + Capmatinib | Part II: Encorafenib + Binimetinib + Buparlisib
Number analyzed (Participants) | 38 | 1 | 13 | 6
Participants
  Encorafenib | 14 | 0 | 4 | 2
  Binimetinib | 13 | 0 | 5 | 3
  Ribociclib: number analyzed (Participants) | 38 | 0 | 0 | 0
  Ribociclib | 11 |  |  |
  Infigratinib: number analyzed (Participants) | 0 | 1 | 0 | 0
  Infigratinib |  | 0 |  |
  Capmatinib: number analyzed (Participants) | 0 | 0 | 13 | 0
  Capmatinib |  |  | 5 |
  Buparlisib: number analyzed (Participants) | 0 | 0 | 0 | 6
  Buparlisib |  |  |  | 2

15. Secondary Outcome: Number of Participants With At Least One Dose Reduction: Part I
Description: In this outcome measure number of participants with at least 1 dose reduction for encorafenib and binimetinib were reported.
Time Frame: During study treatment (maximum treatment exposure for Part I was 403.7 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Encorafenib + Binimetinib (Naive) | Part I: Encorafenib + Binimetinib (Non-naive)
Number analyzed (Participants) | 75 | 83
Participants
  Encorafenib | 9 | 14
  Binimetinib | 32 | 28

16. Secondary Outcome: Number of Participants With At Least One Dose Reduction: Part II
Description: In this outcome measure number of participants with at least 1 dose reduction for encorafenib, binimetinib, and each third combination agent were reported.
Time Frame: During study treatment (maximum treatment exposure for Part II was 97.0 weeks)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Part II: Encorafenib + Binimetinib + Ribociclib | Part II: Encorafenib + Binimetinib + Infigratinib | Part II: Encorafenib + Binimetinib + Capmatinib | Part II: Encorafenib + Binimetinib + Buparlisib
Number analyzed (Participants) | 38 | 1 | 13 | 6
Participants
  Encorafenib | 1 | 0 | 0 | 1
  Binimetinib | 11 | 0 | 5 | 3
  Ribociclib: number analyzed (Participants) | 38 | 0 | 0 | 0
  Ribociclib | 1 |  |  |
  Infigratinib: number analyzed (Participants) | 0 | 1 | 0 | 0
  Infigratinib |  | 0 |  |
  Capmatinib: number analyzed (Participants) | 0 | 0 | 13 | 0
  Capmatinib |  |  | 7 |
  Buparlisib: number analyzed (Participants) | 0 | 0 | 0 | 6
  Buparlisib |  |  |  | 1

17. Secondary Outcome: Actual Dose Intensity: Part I
Description: Dose intensity across all cycles = cumulative dose/duration of exposure. Treatment cycle for encorafenib and binimetinib =21 days.
Time Frame: During study treatment (maximum treatment exposure for Part I was 403.7 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Milligram per day
Arm/Group | Part I: Encorafenib + Binimetinib (Naive) | Part I: Encorafenib + Binimetinib (Non-naive)
Number analyzed (Participants) | 75 | 83
Milligram per day
  Encorafenib | 425.311 (53.5392) | 408.711 (65.5297)
  Binimetinib | 81.920 (13.0994) | 82.083 (10.9117)

18. Secondary Outcome: Actual Dose Intensity: Part II
Description: Dose intensity = cumulative dose/ duration of exposure. Treatment cycle = 21days for the combination treatment with buparlisib and capmatinib and 28 days for the combination treatment with ribociclib and infigratinib.
Time Frame: During study treatment (maximum treatment exposure for Part II was 97.0 weeks)
Population: Safety set included all participants who received at least 1 dose of 3rd combination agent for Part II and had at least 1 valid post-baseline safety assessment. Here, "Number Analyzed" signifies number of participants evaluable for specified drug.
Measure: Mean (Standard Deviation); unit: Milligram per day
Arm/Group | Part II: Encorafenib + Binimetinib + Ribociclib | Part II: Encorafenib + Binimetinib + Infigratinib | Part II: Encorafenib + Binimetinib + Capmatinib | Part II: Encorafenib + Binimetinib + Buparlisib
Number analyzed (Participants) | 38 | 1 | 13 | 6
Milligram per day
  Encorafenib | 197.856 (42.6637) | 450.000 (NA) — Only 1 participant evaluable. | 195.945 (8.4015) | 405.014 (102.5218)
  Binimetinib | 79.749 (14.7267) | 90.000 (NA) — Only 1 participant evaluable. | 87.373 (3.6593) | 78.791 (20.1538)
  Ribociclib: number analyzed (Participants) | 38 | 0 | 0 | 0
  Ribociclib | 486.628 (79.4485) |  |  |
  Infigratinib: number analyzed (Participants) | 0 | 1 | 0 | 0
  Infigratinib |  | 60.227 (NA) — Only 1 participant evaluable. |  |
  Capmatinib: number analyzed (Participants) | 0 | 0 | 13 | 0
  Capmatinib |  |  | 579.519 (259.1157) |
  Buparlisib: number analyzed (Participants) | 0 | 0 | 0 | 6
  Buparlisib |  |  |  | 72.206 (15.7019)

19. Secondary Outcome: Progression-Free Survival (PFS): Part I
Description: PFS was defined as the time from the start date of study drug in Part I until documented PD or death due to any cause. All participants who had not progressed or died at the time of the data cut-off were censored at the date of last tumor assessment (other than those who were unknown or missing) prior to cut-off date or start date of new anti-neoplastic therapy, whichever is earlier. Per RECIST 1.1, PD= At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Kaplan Meier method used for estimation.
Time Frame: From start of study drug until documented PD or death due to any cause or censoring date (maximum treatment exposure for Part I was 403.7 weeks)
Population: For Part I, FAS consisted of all participants who received at least 1 dose (partial or full) of encorafenib or binimetinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part I: Encorafenib + Binimetinib (Naive) | Part I: Encorafenib + Binimetinib (Non-naive)
Number analyzed (Participants) | 75 | 83
Months | 11.1 [8.1 to 15.0] | 3.3 [2.1 to 4.7]

20. Secondary Outcome: PFS: Part II
Description: PFS was defined as the time from the start date of study drug in Part II until documented PD or death due to any cause. All participants who had not progressed or died at the time of the data cut-off were censored at the date of last tumor assessment (other than those who were unknown or missing) prior to cut-off date or start date of new anti-neoplastic therapy, whichever is earlier. Per RECIST 1.1, PD= At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Kaplan Meier method used for estimation.
Time Frame: From start of study drug until documented PD or death due to any cause or censoring date (maximum treatment exposure for Part II was 97.0 weeks)
Population: For Part II, FAS consisted of all participants who received at least 1 dose of encorafenib or binimetinib or the assigned third agent following the assignment of the triple combination treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part II: Encorafenib + Binimetinib + Ribociclib | Part II: Encorafenib + Binimetinib + Infigratinib | Part II: Encorafenib + Binimetinib + Capmatinib | Part II: Encorafenib + Binimetinib + Buparlisib
Number analyzed (Participants) | 38 | 1 | 13 | 6
Months | 2.1 [1.7 to 2.1] | 2.1 [NA to NA] — Only 1 participant evaluable. | 2.1 [1.0 to 3.7] | 1.4 [0.4 to NA] — Upper limit of 95% CI could not be estimated as there were insufficient number of participants with events.

21. Secondary Outcome: Duration of Response (DOR): Part I
Description: DOR: time between date of first documented response (CR or PR) and date of first documented progression or death due to underlying cancer. If there was no progression or death due to underlying cancer, then the participant was censored at the date of last tumor assessment other than unknown. RECIST v1.1: CR = disappearance of all non-nodal target lesions. Any pathological lymph nodes assigned as target lesions must had a reduction in short axis to <10 mm. Disappearance of all non-target lesions. All lymph nodes assigned a non-target lesion must be non-pathological in size (<10 mm short axis); b) PR = at least a 30% decrease in sum of diameter of all target lesions, taking as reference baseline sum of diameters; c) PD= At least a 20% increase in sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition, sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From date of first documented response (CR or PR) till the date of first documented progression or death due to underlying cancer or censoring date (maximum treatment exposure for Part I was 403.7 weeks)
Population: For Part I, FAS consisted of all participants who received at least 1 dose (partial or full) of encorafenib or binimetinib. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure who were confirmed responders. Kaplan Meier method used for estimation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part I: Encorafenib + Binimetinib (Naive) | Part I: Encorafenib + Binimetinib (Non-naive)
Number analyzed (Participants) | 55 | 21
Months | 10.9 [8.1 to 14.1] | 5.6 [3.9 to 13.0]

22. Secondary Outcome: DOR: Part II
Description: as for outcome 21
Time Frame: From date of first documented response (CR or PR) till the date of first documented progression or death due to underlying cancer or censoring date (maximum treatment exposure for Part II was 97.0 weeks)
Population: For Part II, FAS consisted of all participants who received at least 1 dose of encorafenib or binimetinib or the assigned third agent following the assignment of the triple combination treatment. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure who were confirmed responders. Kaplan Meier method used for estimation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part II: Encorafenib + Binimetinib + Ribociclib | Part II: Encorafenib + Binimetinib + Infigratinib | Part II: Encorafenib + Binimetinib + Capmatinib | Part II: Encorafenib + Binimetinib + Buparlisib
Number analyzed (Participants) | 1 | 0 | 0 | 0
Months | 2.1 [NA to NA] — Only 1 participant was evaluable. |  |  |

23. Secondary Outcome: Time to Response (TTR): Part I
Description: TTR was defined as the time between the start date of study drug in Part I and first documented response (CR or PR). RECIST v1.1: a) CR = disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must had a reduction in short axis to <10 mm. Disappearance of all non-target lesions. In addition, all lymph nodes assigned a non-target lesion must be non-pathological in size (<10 mm short axis) and b) PR = at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. Kaplan Meier method used for estimation.
Time Frame: From start date of study drug till first documented response (CR or PR) (maximum treatment exposure for Part I was 403.7 weeks)
Population: For Part I, FAS consisted of all participants who received at least 1 dose (partial or full) of encorafenib or binimetinib. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure who were responders.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part I: Encorafenib + Binimetinib (Naive) | Part I: Encorafenib + Binimetinib (Non-naive)
Number analyzed (Participants) | 52 | 16
Months | 1.4 [1.38 to 1.41] | 0.72 [0.72 to 0.82]

24. Secondary Outcome: TTR: Part II
Description: TTR was defined as the time between the start date of study drug in Part II and first documented response (CR or PR). RECIST v1.1: a) CR = disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must had a reduction in short axis to <10 mm. Disappearance of all non-target lesions. In addition, all lymph nodes assigned a non-target lesion must be non-pathological in size (<10 mm short axis) and b) PR = at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. Kaplan Meier method used for estimation.
Time Frame: From start date of study drug till first documented response (CR or PR) (maximum treatment exposure for Part II was 97.0 weeks)
Population: For Part II, FAS consisted of all participants who received at least 1 dose of encorafenib or binimetinib or the assigned third agent following the assignment of the triple combination treatment. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure who were responders.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part II: Encorafenib + Binimetinib + Ribociclib | Part II: Encorafenib + Binimetinib + Infigratinib | Part II: Encorafenib + Binimetinib + Capmatinib | Part II: Encorafenib + Binimetinib + Buparlisib
Number analyzed (Participants) | 1 | 0 | 0 | 0
Months | 4.1 [NA to NA] — Only 1 participant was evaluable. |  |  |

25. Secondary Outcome: Disease Control Rate (DCR): Part I
Description: DCR was defined as percentage of participants with a best overall response of CR or PR or SD. RECIST v1.1: a) CR = disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must had a reduction in short axis to <10 mm. Disappearance of all non-target lesions. In addition, all lymph nodes assigned a non-target lesion must be non-pathological in size (<10 mm short axis); b) PR = at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters and c) SD = neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD. PD= At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From start date of study drug till first documented response (CR or PR or SD) (maximum treatment exposure for Part I was 403.7 weeks)
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part I: Encorafenib + Binimetinib (Naive) | Part I: Encorafenib + Binimetinib (Non-naive)
Number analyzed (Participants) | 75 | 83
Percentage of participants | 92.0 [83.4 to 97.0] | 42.2 [31.4 to 53.5]

26. Secondary Outcome: DCR: Part II
Description: as for outcome 25
Time Frame: From start date of study drug till first documented response (CR or PR or SD) (maximum treatment exposure for Part II was 97.0 weeks)
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part II: Encorafenib + Binimetinib + Ribociclib | Part II: Encorafenib + Binimetinib + Infigratinib | Part II: Encorafenib + Binimetinib + Capmatinib | Part II: Encorafenib + Binimetinib + Buparlisib
Number analyzed (Participants) | 38 | 1 | 13 | 6
Percentage of participants | 26.3 [13.4 to 43.1] | 0 [NA to NA] — Only 1 participant was evaluable. | 15.4 [1.9 to 45.4] | 16.7 [0.4 to 64.1]

27. Secondary Outcome: Overall Survival (OS): Part II
Description: OS was defined as the time from the start date of study treatment (3rd agent combined with encorafenib and binimetinib) to date of death due to any cause. If a participant was not known to have died, survival was censored at the date of last known date participant alive. Kaplan Meier method used for estimation.
Time Frame: From date of start of treatment to date of death due to any cause or censoring date (maximum treatment exposure for Part II was 97.0 weeks)
Population: as for outcome 20
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part II: Encorafenib + Binimetinib + Ribociclib | Part II: Encorafenib + Binimetinib + Infigratinib | Part II: Encorafenib + Binimetinib + Capmatinib | Part II: Encorafenib + Binimetinib + Buparlisib
Number analyzed (Participants) | 38 | 1 | 13 | 6
Months | 10.4 [6.0 to 16.7] | 20.8 [NA to NA] — Only 1 participant was evaluable. | 5.6 [1.7 to NA] — Upper limit was not estimable due to insufficient number of participants with events. | 2.5 [0.4 to NA] — Upper limit was not estimable due to insufficient number of participants with events.

28. Secondary Outcome: Summary of Genomic Biomarkers From Tumor Samples: Part I
Description: Number of participants with multiple alterations in genomic biomarkers like biomarker BRAF, CCND1, CDK4, EGFR, FGFR1, FGFR4, KRAS, MET, NRAS, PIK3CA, and PTEN were reported and alterations included copy number variant/copy number ratio (CNV/CNR), rearrangement, short variant. It was not necessary that all biomarkers had all alterations. Baseline = last non-missing value prior to the first dose of study treatment.
Time Frame: Baseline up to end of treatment (EOT) (maximum treatment exposure for Part I was 403.7 weeks)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Encorafenib + Binimetinib (Naive) | Part I: Encorafenib + Binimetinib (Non-naive)
Number analyzed (Participants) | 75 | 83
Participants
  BRAF: CNV/CNR at Baseline | 4 | 9
  BRAF: CNV/CNR at EOT | 2 | 3
  BRAF: Rearrangement/Genomic Position at Baseline chr7:140482508-140482692 | 0 | 1
  BRAF: Rearrangement/Genomic Position at Baseline chr7:140487121-140487285 | 0 | 1
  BRAF: Rearrangement/Genomic Position at Baseline chr7:140487916-140488167 | 0 | 1
  BRAF: Rearrangement/Genomic Position at Baseline chr7:140488878-140489055 | 0 | 1
  BRAF: Rearrangement/Genomic Position at Baseline cchr7:140489413-140489576 | 0 | 1
  BRAF: Rearrangement/Genomic Position at Baseline chr7:140490446-140490656 | 0 | 1
  BRAF: Rearrangement/Genomic Position at Baseline chr7:140491528-140491878 | 0 | 1
  BRAF: Rearrangement/Genomic Position at Baseline chr7:140491580-140491878 | 0 | 1
  BRAF: Rearrangement/Genomic Position at Baseline chr7:140492969-140493301 | 0 | 1
  BRAF: Rearrangement/Genomic Position at EOT chr7:140481691-140482150 | 1 | 0
  BRAF: Rearrangement/Genomic Position at EOT chr7:140482057-140482467 | 0 | 1
  BRAF: Rearrangement/Genomic Position at EOT chr7:140482081-140482482 | 1 | 0
  BRAF: Rearrangement/Genomic Position at EOT chr7:140482088-140482296 | 0 | 1
  BRAF: Rearrangement/Genomic Position at EOT chr7:140482167-140482382 | 1 | 0
  BRAF: Rearrangement/Genomic Position at EOT chr7:140482495-140482731 | 0 | 1
  BRAF: Rearrangement/Genomic Position at EOT chr7:140482644-140482867 | 0 | 1
  BRAF: Rearrangement/Genomic Position at EOT chr7:140483058-140483257 | 1 | 0
  BRAF: Rearrangement/Genomic Position at EOT chr7:140486136-140486408 | 1 | 0
  BRAF: Rearrangement/Genomic Position at EOT chr7:140486274-140486561 | 0 | 1
  BRAF: Rearrangement/Genomic Position at EOT chr7:140489019-140489575 | 0 | 1
  BRAF: Rearrangement/Genomic Position at EOT chr7:140489219-140489431 | 1 | 0
  BRAF: Rearrangement/Genomic Position at EOT chr7:140489830-140490002 | 0 | 1
  BRAF: Rearrangement/Genomic Position at EOT chr7:140491411-140491879 | 0 | 1
  BRAF: Rearrangement/Genomic Position at EOT chr7:140492091-140492240 | 1 | 0
  BRAF: Rearrangement/Genomic Position at EOT chr7:140492379-140492708 | 0 | 1
  BRAF: Rearrangement/Genomic Position at EOT chr7:140492714-140492997 | 0 | 1
  BRAF: Rearrangement/Genomic Position at EOT chr7:140493601-140493951 | 0 | 1
  BRAF: Rearrangement/Genomic Position at EOT chr7:140493858-140494232 | 1 | 0
  BRAF: Short variant/amino acid change at Baseline V600E | 46 | 53
  BRAF: Short variant/amino acid change at Baseline V600G | 1 | 0
  BRAF: Short variant/amino acid change at Baseline V600K | 4 | 7
  BRAF: Short variant/amino acid change at Baseline V600R | 1 | 0
  BRAF: Short variant/amino acid change at EOT V600E | 18 | 19
  BRAF: Short variant/amino acid change at EOT V600K | 0 | 4
  BRAF: Short variant/amino acid change at EOT V600R | 1 | 0
  CCND1: CNV/CNR at Baseline | 1 | 0
  CDK4: CNV/CNR at Baseline | 3 | 2
  EGFR: CNV/CNR at Baseline | 1 | 3
  EGFR: CNV/CNR at EOT | 1 | 1
  FGFR1: CNV/CNR at Baseline | 1 | 0
  FGFR1: CNV/CNR at EOT | 1 | 0
  FGFR4: CNV/CNR at Baseline | 1 | 0
  KRAS: CNV/CNR at Baseline | 2 | 0
  MET: CNV/CNR at Baseline | 4 | 6
  MET: CNV/CNR at EOT | 3 | 5
  MET: Rearrangement/Genomic Position at EOT chr7:116321020-116321260 | 1 | 0
  NRAS: CNV/CNR at Baseline | 0 | 1
  PIK3CA: CNV/CNR at Baseline | 1 | 0
  PTEN: CNV/CNR at Baseline | 4 | 13
  PTEN: CNV/CNR at EOT | 5 | 10
  PTEN: Rearrangement/Genomic Position at EOT chr10:89720538-89720776 | 0 | 1

29. Secondary Outcome: Plasma Concentration for Encorafenib (LGX): Part I
Description: In results reported below, following abbreviation have been used: Cycle 1 (C1), Day 1 (D1), Day 8 (D8), Day 15 (D15), Day 21 (D21), Cycle 2 (C2), Cycle 3 (C3), Cycle 4 (C4), Cycle 5 (C5) and end of treatment (EOT). Maximum treatment exposure for Part I was of 403.7 weeks.
Time Frame: C1 (1.5 hrs post-dose on D1; pre-dose, 1.5 hrs post-dose on D15); C2 (pre-dose on D8 and D21); C3 pre-dose on D15; C4 pre-dose on D15; C5 pre-dose on D15; EOT
Population: Pharmacokinetic analysis set (PAS) consisted of all participants who had at least one blood sample providing evaluable pharmacokinetic (PK) data. All participants reported under "Number of Participants Analyzed" contributed data to the table but may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable for specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part I: Encorafenib + Binimetinib (Naive) | Part I: Encorafenib + Binimetinib (Non-naive)
Number analyzed (Participants) | 75 | 78
Nanogram per milliliter
  C1 D1, 1.5 hr: number analyzed (Participants) | 59 | 55
  C1 D1, 1.5 hr | 4820 (114.2) | 4480 (124.4)
  C1 D15, Pre-dose: number analyzed (Participants) | 68 | 59
  C1 D15, Pre-dose | 10.0 (81.6) | 13.8 (104.4)
  C1 D15, 1.5 hr: number analyzed (Participants) | 52 | 54
  C1 D15, 1.5 hr | 2470 (116.7) | 2910 (91.6)
  C2 D8, Pre-dose: number analyzed (Participants) | 69 | 48
  C2 D8, Pre-dose | 9.96 (81.7) | 14.7 (117.5)
  C2 D21, Pre-dose: number analyzed (Participants) | 62 | 41
  C2 D21, Pre-dose | 9.04 (84.2) | 15.6 (156.3)
  C3 D15, Pre-dose: number analyzed (Participants) | 68 | 41
  C3 D15, Pre-dose | 8.43 (82.3) | 11.2 (114.3)
  C4 D15, Pre-dose: number analyzed (Participants) | 63 | 30
  C4 D15, Pre-dose | 9.21 (100.3) | 12.3 (108.9)
  C5 D15, Pre-dose: number analyzed (Participants) | 56 | 30
  C5 D15, Pre-dose | 8.84 (59.4) | 11.9 (72.7)
  EOT: number analyzed (Participants) | 35 | 47
  EOT | 19.6 (399.9) | 34.5 (890.3)

30. Secondary Outcome: Plasma Concentration for Encorafenib (LGX): Part II
Description: In results reported below, following abbreviation have been used: Cycle 1 (C1), Day 1 (D1), Day 8 (D8), Day 15 (D15), Day 16 (D16), Day 21 (D21), Cycle 2 (C2), Cycle 3 (C3), Cycle 4 (C4), Cycle 5 (C5). Maximum treatment exposure for Part II was of 97.0 weeks.
Time Frame: C1 (1.5, 4 hrs post-dose on D1; pre-dose on D8; pre-dose, 0.5, 1.5, 2.5, 4, 6, 8 hrs post-dose on D15; 24 hrs post-dose on D16; pre-dose on D21); C2 (pre-dose on D1 and D15); C3 pre-dose on D1; C4 pre-dose on D1; C5 pre-dose on D1; EOT
Population: PAS consisted of all participants who had at least one blood sample providing evaluable PK data. All participants reported under "Number of Participants Analyzed" contributed data to the table but may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable for specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 60 mg: Participants received encorafenib 450 mg once a day and binimetinib 45 mg twice a day along with buparlisib 60 mg once a day.
- Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 90 mg: Participants received encorafenib 450 mg once a day and binimetinib 45 mg twice a day along with buparlisib 90 mg once a day.
- Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Infigratinib 75 mg: Participants received encorafenib 450 mg once a day and binimetinib 45 mg twice a day along with infigratinib 75 mg once a day.
- Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 200 mg: Participants received encorafenib 200 mg once a day and binimetinib 45 mg twice a day along with capmatinib 200 mg twice a day.
- Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 300 mg: Participants received encorafenib 200 mg once a day and binimetinib 45 mg twice a day along with capmatinib 300 mg twice a day.
- Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 400 mg: Participants received encorafenib 200 mg once a day and binimetinib 45 mg twice a day along with capmatinib 400 mg twice a day.
- Part II: Encorafenib 100 mg/ Binimetinib 30 mg + Ribociclib 600 mg: Participants received encorafenib 100 mg once a day and binimetinib 30 mg twice a day along with ribociclib 600 mg once a day.
- Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 400 mg: Participants received encorafenib 200 mg once a day and binimetinib 30 mg twice a day along with ribociclib 400 mg once a day.
- Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 600 mg: Participants received encorafenib 200 mg once a day and binimetinib 30 mg twice a day along with ribociclib 600 mg once a day.
- Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 400 mg: Participants received encorafenib 200 mg once a day and binimetinib 45 mg twice a day along with ribociclib 400 mg once a day.
- Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 600 mg: Participants received encorafenib 200 mg once a day and binimetinib 45 mg twice a day along with ribociclib 600 mg once a day.
Arm/Group | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 60 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 90 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Infigratinib 75 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 200 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 300 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 400 mg | Part II: Encorafenib 100 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 600 mg
Number analyzed (Participants) | 3 | 3 | 1 | 5 | 1 | 5 | 1 | 1 | 3 | 1 | 29
Nanogram per milliliter
  C1 D1: 1.5 hrs: number analyzed (Participants) | 0 | 2 | 1 | 2 | 1 | 3 | 1 | 1 | 2 | 0 | 22
  C1 D1: 1.5 hrs |  | 3430 (17.6) | 1860 (NA) — Only 1 participant evaluable. | 1130 (3.8) | 3750 (NA) — Only 1 participant evaluable. | 1770 (62.9) | 878 (NA) — Only 1 participant evaluable. | 2030 (NA) — Only 1 participant evaluable. | 847 (28.1) |  | 1600 (85.6)
  C1 D1: 4 hrs: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 24
  C1 D1: 4 hrs |  |  |  |  |  |  | 238 (NA) — Only 1 participant evaluable. | 297 (NA) — Only 1 participant evaluable. | 626 (65.7) |  | 596 (51.1)
  C1 D8: Pre-dose: number analyzed (Participants) | 3 | 2 | 1 | 3 | 1 | 4 | 1 | 1 | 2 | 1 | 23
  C1 D8: Pre-dose | 8.97 (89.0) | 21.3 (150.6) | 12.4 (NA) — Only 1 participant evaluable. | 10.3 (54.4) | 6.21 (NA) — Only 1 participant evaluable. | 11.7 (56.4) | 12.5 (NA) — Only 1 participant evaluable. | 15.2 (NA) — Only 1 participant evaluable. | 9.39 (15.9) | 7.15 (NA) — Only 1 participant evaluable. | 16.2 (116.1)
  C1 D15: Pre-dose: number analyzed (Participants) | 3 | 2 | 1 | 4 | 1 | 4 | 1 | 1 | 2 | 0 | 22
  C1 D15: Pre-dose | 11.2 (106.3) | 18.6 (159.4) | 7.74 (NA) — Only 1 participant evaluable. | 9.95 (40.1) | 7.95 (NA) — Only 1 participant evaluable. | 13.5 (35.0) | 9.28 (NA) — Only 1 participant evaluable. | 10.3 (NA) — Only 1 participant evaluable. | 7.75 (37.3) |  | 20.9 (188.5)
  C1 D15: 0.5 hr: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 0 | 22
  C1 D15: 0.5 hr | 437 (228.2) | 625 (19.5) | 1690 (NA) — Only 1 participant evaluable. | 262 (345.5) | 139 (NA) — Only 1 participant evaluable. | 127 (216.1) | 8.55 (NA) — Only 1 participant evaluable. | 601 (NA) — Only 1 participant evaluable. | 473 (1248.5) |  | 175 (252.7)
  C1 D15: 1.5 hrs: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 0 | 22
  C1 D15: 1.5 hrs | 3050 (59.6) | 2150 (54.6) | 2100 (NA) — Only 1 participant evaluable. | 1550 (62.4) | 2890 (NA) — Only 1 participant evaluable. | 2500 (27.9) | 366 (NA) — Only 1 participant evaluable. | 1960 (NA) — Only 1 participant evaluable. | 1450 (3.9) |  | 1850 (69.7)
  C1 D15: 2.5 hrs: number analyzed (Participants) | 3 | 2 | 1 | 5 | 0 | 4 | 1 | 1 | 1 | 0 | 22
  C1 D15: 2.5 hrs | 1420 (39.6) | 1320 (30.0) | 1020 (NA) — Only 1 participant evaluable. | 808 (55.0) |  | 1550 (34.4) | 622 (NA) — Only 1 participant evaluable. | 981 (NA) — Only 1 participant evaluable. | 686 (NA) — Only 1 participant evaluable. |  | 1510 (48.2)
  C1 D15: 4 hrs: number analyzed (Participants) | 3 | 2 | 1 | 4 | 1 | 4 | 1 | 0 | 2 | 0 | 23
  C1 D15: 4 hrs | 649 (37.5) | 770 (6.2) | 397 (NA) — Only 1 participant evaluable. | 453 (24.3) | 1160 (NA) — Only 1 participant evaluable. | 667 (20.4) | 389 (NA) — Only 1 participant evaluable. |  | 478 (39.6) |  | 1020 (34.3)
  C1 D15: 6 hrs: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 0 | 19
  C1 D15: 6 hrs | 246 (94.6) | 433 (45.0) | 211 (NA) — Only 1 participant evaluable. | 165 (68.8) | 266 (NA) — Only 1 participant evaluable. | 317 (26.8) | 209 (NA) — Only 1 participant evaluable. | 199 (NA) — Only 1 participant evaluable. | 203 (11.1) |  | 567 (51.5)
  C1 D15: 8 hrs: number analyzed (Participants) | 3 | 2 | 0 | 5 | 1 | 3 | 1 | 1 | 2 | 0 | 20
  C1 D15: 8 hrs | 180 (94.5) | 276 (103.8) |  | 115 (55.4) | 257 (NA) — Only 1 participant evaluable. | 217 (34.5) | 142 (NA) — Only 1 participant evaluable. | 132 (NA) — Only 1 participant evaluable. | 109 (2.6) |  | 412 (62.3)
  C1 D16: 24 hrs: number analyzed (Participants) | 3 | 2 | 1 | 4 | 1 | 4 | 1 | 1 | 2 | 0 | 24
  C1 D16: 24 hrs | 11.3 (45.3) | 25.1 (2066.8) | 6.76 (NA) — Only 1 participant evaluable. | 8.10 (43.1) | 5.20 (NA) — Only 1 participant evaluable. | 15.0 (20.9) | 10.7 (NA) — Only 1 participant evaluable. | 7.85 (NA) — Only 1 participant evaluable. | 10.8 (106.1) |  | 22.8 (199.0)
  C1 D21: Pre-dose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 20
  C1 D21: Pre-dose |  |  | 10.4 (NA) — Only 1 participant evaluable. |  |  |  | 13.6 (NA) — Only 1 participant evaluable. | 13.9 (NA) — Only 1 participant evaluable. | 12.4 (60.4) | 20.3 (NA) — Only 1 participant evaluable. | 17.5 (106.4)
  C2 D1: Pre-dose: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 3 | 1 | 1 | 2 | 1 | 18
  C2 D1: Pre-dose | 13.5 (193.0) | 32.6 (202.9) | 12.7 (NA) — Only 1 participant evaluable. | 19.9 (210.5) | 2.91 (NA) — Only 1 participant evaluable. | 14.0 (30.3) | 8.50 (NA) — Only 1 participant evaluable. | 82.5 (NA) — Only 1 participant evaluable. | 8.19 (42.2) | 19.2 (NA) — Only 1 participant evaluable. | 11.9 (100.9)
  C2 D15: Pre-dose: number analyzed (Participants) | 1 | 1 | 1 | 4 | 0 | 4 | 1 | 1 | 2 | 1 | 14
  C2 D15: Pre-dose | 41.3 (NA) — Only 1 participant evaluable. | 15.6 (NA) — Only 1 participant evaluable. | 13.9 (NA) — Only 1 participant evaluable. | 9.68 (36.5) |  | 8.49 (70.5) | 11.1 (NA) — Only 1 participant evaluable. | 16.5 (NA) — Only 1 participant evaluable. | 12.3 (24.3) | 8.95 (NA) — Only 1 participant evaluable. | 21.3 (115.3)
  C3 D1: Pre-dose: number analyzed (Participants) | 1 | 0 | 1 | 2 | 0 | 4 | 0 | 1 | 0 | 0 | 15
  C3 D1: Pre-dose | 13.9 (NA) — Only 1 participant evaluable. |  | 20.5 (NA) — Only 1 participant evaluable. | 23.2 (33.1) |  | 10.1 (72.1) |  | NA (NA) — Participant had below limit of the quantitation (BLQ) value. |  |  | 9.34 (125.7)
  C4 D1: Pre-dose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 6
  C4 D1: Pre-dose | 30.2 (NA) — Only 1 participant evaluable. |  |  |  |  | 12.5 (11.4) | 5.95 (NA) — Only 1 participant evaluable. | 7.28 (NA) — Only 1 participant evaluable. |  |  | 13.1 (21.8)
  C5 D1: Pre-dose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 5
  C5 D1: Pre-dose | 749 (NA) — Only 1 participant evaluable. |  |  |  |  |  | 10.7 (NA) — Only 1 participant evaluable. | 9.84 (NA) — Only 1 participant evaluable. |  |  | 9.15 (44.0)
  EOT: number analyzed (Participants) | 2 | 1 | 1 | 3 | 1 | 4 | 1 | 1 | 2 | 1 | 22
  EOT | 1.77 (NA) — Out of 2, 1 participant had BLQ value. | NA (NA) — Participant had BLQ value. | 14.3 (NA) — Only 1 participant evaluable. | NA (NA) — All participants had BLQ value. | NA (NA) — Participant had BLQ value. | 13.9 (66.6) | 8.24 (NA) — Only 1 participant evaluable. | 6.81 (NA) — Only 1 participant evaluable. | 24.5 (259.8) | NA (NA) — Participant had BLQ value. | 16.6 (265.0)

31. Secondary Outcome: Plasma Concentration for Binimetinib (MEK) and Its Metabolite: Part I
Description: AR00426032 is metabolite of binimetinib. Maximum treatment exposure for Part I was of 403.7 weeks.
Time Frame: as for outcome 29
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part I: Encorafenib + Binimetinib (Naive) | Part I: Encorafenib + Binimetinib (Non-naive)
Number analyzed (Participants) | 75 | 78
Nanogram per milliliter
  Binimetinib: C1 D1, 1.5 hr: number analyzed (Participants) | 58 | 60
  Binimetinib: C1 D1, 1.5 hr | 551 (88.8) | 482 (73.4)
  Binimetinib: C1 D15, Pre-dose: number analyzed (Participants) | 66 | 56
  Binimetinib: C1 D15, Pre-dose | 40.3 (63.5) | 43.3 (72.9)
  Binimetinib: C1 D15, 1.5 hr: number analyzed (Participants) | 53 | 54
  Binimetinib: C1 D15, 1.5 hr | 461 (70.2) | 451 (50.2)
  Binimetinib: C2 D8, Pre-dose: number analyzed (Participants) | 69 | 46
  Binimetinib: C2 D8, Pre-dose | 39.9 (58.8) | 44.8 (73.0)
  Binimetinib: C2 D21, Pre-dose: number analyzed (Participants) | 62 | 39
  Binimetinib: C2 D21, Pre-dose | 38.9 (54.9) | 53.1 (78.2)
  Binimetinib: C3 D15, Pre-dose: number analyzed (Participants) | 65 | 41
  Binimetinib: C3 D15, Pre-dose | 41.9 (60.4) | 38.7 (94.6)
  Binimetinib: C4 D15, Pre-dose: number analyzed (Participants) | 61 | 30
  Binimetinib: C4 D15, Pre-dose | 36.2 (68.6) | 38.8 (57.4)
  Binimetinib: C5 D15, Pre-dose: number analyzed (Participants) | 56 | 30
  Binimetinib: C5 D15, Pre-dose | 41.3 (55.7) | 39.2 (76.1)
  Binimetinib: EOT: number analyzed (Participants) | 35 | 47
  Binimetinib: EOT | 33.2 (179.4) | 52.8 (180.4)
  AR00426032: C1 D1, 1.5 hr: number analyzed (Participants) | 58 | 60
  AR00426032: C1 D1, 1.5 hr | 57.6 (93.5) | 47.5 (101.6)
  AR00426032: C1 D15, Pre-dose: number analyzed (Participants) | 66 | 56
  AR00426032: C1 D15, Pre-dose | 4.13 (70.8) | 4.50 (64.0)
  AR00426032: C1 D15, 1.5 hr: number analyzed (Participants) | 52 | 54
  AR00426032: C1 D15, 1.5 hr | 30.6 (110.9) | 31.9 (84.0)
  AR00426032: C2 D8, Pre-dose: number analyzed (Participants) | 69 | 46
  AR00426032: C2 D8, Pre-dose | 3.63 (60.2) | 4.17 (88.1)
  AR00426032: C2 D21, Pre-dose: number analyzed (Participants) | 62 | 39
  AR00426032: C2 D21, Pre-dose | 4.11 (61.0) | 4.39 (80.2)
  AR00426032: C3 D15, Pre-dose: number analyzed (Participants) | 64 | 41
  AR00426032: C3 D15, Pre-dose | 3.71 (59.5) | 3.90 (60.6)
  AR00426032: C4 D15, Pre-dose: number analyzed (Participants) | 61 | 30
  AR00426032: C4 D15, Pre-dose | 3.48 (65.8) | 3.81 (56.9)
  AR00426032: C5 D15, Pre-dose: number analyzed (Participants) | 56 | 30
  AR00426032: C5 D15, Pre-dose | 3.77 (66.9) | 3.36 (67.3)
  AR00426032: EOT: number analyzed (Participants) | 33 | 47
  AR00426032: EOT | 4.09 (90.8) | 5.88 (118.0)

32. Secondary Outcome: Plasma Concentration for Binimetinib (MEK) and Its Metabolite: Part II
Description: AR00426032 is metabolite of binimetinib. Maximum treatment exposure for Part II was of 97.0 weeks.
Time Frame: as for outcome 30
Population: PAS consisted of all participants who had at least one blood sample providing evaluable PK data. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable for specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 60 mg: Participants received encorafenib 450 mg once in a day (QD) and binimetinib 45 mg twice in a day (BID) and buparlisib 60 mg QD.
- Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 90 mg: Participants received encorafenib 450 mg QD and binimetinib 45 mg BID and buparlisib 90 mg QD.
- Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Infigratinib 75 mg: Participants received encorafenib 450 mg QD and binimetinib 45 mg BID and infigratinib 75 mg QD.
- Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 200 mg: Participants received encorafenib 200 mg QD and binimetinib 45 mg BID and capmatinib 200 mg BID.
- Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 300 mg: Participants received encorafenib 200 mg QD and binimetinib 45 mg BID and capmatinib 300 mg BID.
- Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 400 mg: Participants received encorafenib 200 mg QD and binimetinib 45 mg BID and capmatinib 400 mg BID.
- Part II: Encorafenib 100 mg/ Binimetinib 30 mg + Ribociclib 600 mg: Participants received encorafenib 100 mg QD and binimetinib 30 mg BID and ribociclib 600 mg QD.
- Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 400 mg: Participants received encorafenib 200 mg QD and binimetinib 30 mg BID and ribociclib 400 mg QD.
- Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 600 mg: Participants received encorafenib 200 mg QD and binimetinib 30 mg BID and ribociclib 600 mg QD.
- Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 400 mg: Participants received encorafenib 200 mg QD and binimetinib 45 mg BID and ribociclib 400 mg QD.
- Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 600 mg: Participants received encorafenib 200 mg QD and binimetinib 45 mg BID and ribociclib 600 mg QD.
- Part II: Encorafenib 300 mg/ Binimetinib 30 mg + Ribociclib 600 mg: Participants received encorafenib 300 mg QD and binimetinib 30 mg BID and ribociclib 600 mg QD.
- Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Ribociclib 600 mg: Participants received encorafenib 450 mg QD and binimetinib 45 mg BID and ribociclib 600 mg QD.
Arm/Group | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 60 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 90 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Infigratinib 75 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 200 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 300 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 400 mg | Part II: Encorafenib 100 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 600 mg | Part II: Encorafenib 300 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Ribociclib 600 mg
Number analyzed (Participants) | 3 | 3 | 1 | 5 | 1 | 5 | 1 | 1 | 3 | 1 | 29 | 1 | 1
Nanogram per milliliter
  Binimetinib, C1 D1: 1.5 hrs: number analyzed (Participants) | 0 | 2 | 1 | 2 | 1 | 3 | 1 | 1 | 2 | 0 | 21 | 1 | 1
  Binimetinib, C1 D1: 1.5 hrs |  | 410 (48.8) | 416 (NA) — Only 1 participant evaluable. | 313 (25.6) | 1100 (NA) — Only 1 participant evaluable. | 508 (130.2) | 396 (NA) — Only 1 participant evaluable. | 649 (NA) — Only 1 participant evaluable. | 273 (24.6) |  | 446 (59.8) | 522 (NA) — Only 1 participant evaluable. | 1230 (NA) — Only 1 participant evaluable.
  Binimetinib, C1 D1: 4 hrs: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 24 | 1 | 0
  Binimetinib, C1 D1: 4 hrs |  |  |  |  |  |  | 152 (NA) — Only 1 participant evaluable. | 106 (NA) — Only 1 participant evaluable. | 129 (25.8) |  | 215 (44.5) | 99.5 (NA) — Only 1 participant evaluable. |
  Binimetinib, C1 D8: Pre-dose: number analyzed (Participants) | 3 | 2 | 1 | 3 | 1 | 4 | 1 | 1 | 2 | 1 | 21 | 1 | 0
  Binimetinib, C1 D8: Pre-dose | 41.6 (21.7) | 51.1 (9.7) | 46.0 (NA) — Only 1 participant evaluable. | 74.6 (34.5) | 27.2 (NA) — Only 1 participant evaluable. | 67.4 (63.1) | 63.0 (NA) — Only 1 participant evaluable. | 31.5 (NA) — Only 1 participant evaluable. | 25.1 (1.7) | 27.2 (NA) — Only 1 participant evaluable. | 51.0 (67.8) | 37.3 (NA) — Only 1 participant evaluable. |
  Binimetinib, C1 D15: Pre-dose: number analyzed (Participants) | 3 | 2 | 1 | 4 | 1 | 4 | 1 | 1 | 2 | 0 | 22 | 1 | 0
  Binimetinib, C1 D15: Pre-dose | 32.0 (17.1) | 39.1 (57.4) | 33.9 (NA) — Only 1 participant evaluable. | 85.6 (53.7) | 47.3 (NA) — Only 1 participant evaluable. | 50.9 (34.4) | 54.3 (NA) — Only 1 participant evaluable. | 28.3 (NA) — Only 1 participant evaluable. | 21.1 (23.7) |  | 48.2 (70.0) | 36.2 (NA) — Only 1 participant evaluable. |
  Binimetinib, C1 D15: 0.5 hr: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 0 | 22 | 0 | 0
  Binimetinib, C1 D15: 0.5 hr | 150 (36.1) | 143 (496.2) | 315 (NA) — Only 1 participant evaluable. | 430 (26.8) | 401 (NA) — Only 1 participant evaluable. | 180 (91.5) | 229 (NA) — Only 1 participant evaluable. | 389 (NA) — Only 1 participant evaluable. | 161 (54.7) |  | 158 (90.1) |  |
  Binimetinib, C1 D15: 1.5 hrs: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 0 | 22 | 0 | 0
  Binimetinib, C1 D15: 1.5 hrs | 386 (41.1) | 187 (351.0) | 413 (NA) — Only 1 participant evaluable. | 489 (27.1) | 797 (NA) — Only 1 participant evaluable. | 734 (45.6) | 261 (NA) — Only 1 participant evaluable. | 520 (NA) — Only 1 participant evaluable. | 313 (15.9) |  | 437 (46.5) |  |
  Binimetinib, C1 D15: 2.5 hrs: number analyzed (Participants) | 3 | 2 | 1 | 5 | 0 | 4 | 1 | 1 | 1 | 0 | 22 | 1 | 0
  Binimetinib, C1 D15: 2.5 hrs | 250 (17.1) | 143 (172.4) | 235 (NA) — Only 1 participant evaluable. | 295 (29.7) |  | 491 (38.0) | 207 (NA) — Only 1 participant evaluable. | 331 (NA) — Only 1 participant evaluable. | 154 (NA) — Only 1 participant evaluable. |  | 380 (31.2) | 178 (NA) — Only 1 participant evaluable. |
  Binimetinib, C1 D15: 4 hrs: number analyzed (Participants) | 3 | 2 | 1 | 4 | 1 | 4 | 1 | 0 | 2 | 0 | 23 | 0 | 0
  Binimetinib, C1 D15: 4 hrs | 147 (21.4) | 125 (62.1) | 98.0 (NA) — Only 1 participant evaluable. | 166 (48.9) | 264 (NA) — Only 1 participant evaluable. | 266 (32.5) | 130 (NA) — Only 1 participant evaluable. |  | 98.0 (60.0) |  | 241 (28.6) |  |
  Binimetinib, C1 D15: 6 hrs: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 0 | 20 | 0 | 0
  Binimetinib, C1 D15: 6 hrs | 79.0 (36.1) | 97.3 (32.8) | 55.8 (NA) — Only 1 participant evaluable. | 106 (53.3) | 112 (NA) — Only 1 participant evaluable. | 141 (15.1) | 167 (NA) — Only 1 participant evaluable. | 77.4 (NA) — Only 1 participant evaluable. | 53.3 (36.2) |  | 134 (46.5) |  |
  Binimetinib, C1 D15: 8 hrs: number analyzed (Participants) | 3 | 2 | 0 | 5 | 1 | 3 | 1 | 1 | 2 | 0 | 20 | 0 | 0
  Binimetinib, C1 D15: 8 hrs | 74.9 (34.7) | 59.7 (12.6) |  | 107 (40.9) | 132 (NA) — Only 1 participant evaluable. | 102 (12.4) | 116 (NA) — Only 1 participant evaluable | 65.5 (NA) — Only 1 participant evaluable | 42.2 (39.2) |  | 109 (54.8) |  |
  Binimetinib, C1 D16: 24 hrs: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 0 | 23 | 1 | 0
  Binimetinib, C1 D16: 24 hrs | 44.1 (19.1) | 30.2 (59.2) | 42.1 (NA) — Only 1 participant evaluable. | 63.2 (64.0) | 17.6 (NA) — Only 1 participant evaluable. | 55.9 (54.0) | 78.3 (NA) — Only 1 participant evaluable. | 29.8 (NA) — Only 1 participant evaluable. | 23.1 (5.2) |  | 55.2 (66.0) | 40.5 (NA) — Only 1 participant evaluable. |
  Binimetinib, C1 D21: Pre-dose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 19 | 1 | 1
  Binimetinib, C1 D21: Pre-dose |  |  | 34.0 (NA) — Only 1 participant evaluable. |  |  |  | 40.4 (NA) — Only 1 participant evaluable. | 38.8 (NA) — Only 1 participant evaluable. | 13.6 (80.7) | 19.6 (NA) — Only 1 participant evaluable. | 63.2 (51.0) | 35.3 (NA) — Only 1 participant evaluable. | 8.91 (NA) — Only 1 participant evaluable.
  Binimetinib, C2 D1: Pre-dose: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 3 | 1 | 1 | 2 | 1 | 16 | 1 | 1
  Binimetinib, C2 D1: Pre-dose | 38.8 (62.5) | 42.7 (27.8) | 40.5 (NA) — Only 1 participant evaluable. | 118 (120.1) | 24.6 (NA) — Only 1 participant evaluable. | 54.2 (32.4) | 58.3 (NA) — Only 1 participant evaluable. | 174 (NA) — Only 1 participant evaluable. | 23.3 (20.2) | 58.3 (NA) — Only 1 participant evaluable. | 46.0 (71.2) | 22.4 (NA) — Only 1 participant evaluable. | 54.1 (NA) — Only 1 participant evaluable.
  Binimetinib, C2 D15: Pre-dose: number analyzed (Participants) | 1 | 1 | 1 | 4 | 1 | 4 | 1 | 1 | 2 | 1 | 14 | 1 | 1
  Binimetinib, C2 D15: Pre-dose | 63.7 (NA) — Only 1 participant evaluable. | 73.0 (NA) — Only 1 participant evaluable. | 63.9 (NA) — Only 1 participant evaluable. | 40.9 (50.8) | 18.9 (NA) — Only 1 participant evaluable. | 49.8 (21.2) | 63.1 (NA) — Only 1 participant evaluable. | 19.4 (NA) — Only 1 participant evaluable. | 15.2 (18.2) | 14.1 (NA) — Only 1 participant evaluable. | 58.4 (68.3) | 27.3 (NA) — Only 1 participant evaluable. | 34.9 (NA) — Only 1 participant evaluable.
  Binimetinib, C3 D1: Pre-dose: number analyzed (Participants) | 1 | 0 | 1 | 2 | 0 | 4 | 1 | 1 | 0 | 0 | 16 | 1 | 0
  Binimetinib, C3 D1: Pre-dose | 50.0 (NA) — Only 1 participant evaluable. |  | 47.2 (NA) — Only 1 participant evaluable. | 37.8 (189.6) |  | 41.9 (49.0) | 53.4 (NA) — Only 1 participant evaluable. | 4.82 (NA) — Only 1 participant evaluable. |  |  | 45.0 (91.8) | 42.0 (NA) — Only 1 participant evaluable. |
  Binimetinib, C4 D1: Pre-dose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 4 | 0 | 0
  Binimetinib, C4 D1: Pre-dose | 46.1 (NA) — Only 1 participant evaluable. |  |  |  |  | 53.8 (10.6) | 63.6 (NA) — Only 1 participant evaluable. | 40.9 (NA) — Only 1 participant evaluable. |  |  | 77.5 (32.1) |  |
  Binimetinib, C5 D1: Pre-dose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 5 | 0 | 0
  Binimetinib, C5 D1: Pre-dose | 60.0 (NA) — Only 1 participant evaluable. |  |  |  |  |  | 42.3 (NA) — Only 1 participant evaluable. | 28.5 (NA) — Only 1 participant evaluable. |  |  | 73.8 (25.7) |  |
  Binimetinib, EOT: number analyzed (Participants) | 2 | 1 | 1 | 3 | 1 | 4 | 1 | 1 | 2 | 1 | 21 | 0 | 0
  Binimetinib, EOT | NA (NA) — All participants had BLQ value. | NA (NA) — Participant had BLQ value. | 36.3 | NA (NA) — All participants had BLQ value. | NA (NA) — Participant had BLQ value. | 52.1 (18.3) | 41.0 (NA) — Only 1 participant evaluable. | 32.3 (NA) — Only 1 participant evaluable. | 13.8 (205.5) | NA (NA) — Participant had BLQ value. | 29.0 (179.7) |  |
  AR00426032, C1 D1: 1.5 hrs: number analyzed (Participants) | 0 | 2 | 1 | 2 | 0 | 3 | 0 | 1 | 2 | 0 | 21 | 1 | 1
  AR00426032, C1 D1: 1.5 hrs |  | 22.4 (200.6) | 12.9 (NA) — Only 1 participant evaluable. | 11.4 (85.7) |  | 35.9 (274.1) |  | 22.1 (NA) — Only 1 participant evaluable. | 8.05 (68.9) |  | 19.4 (99.3) | 16.3 (NA) — Only 1 participant evaluable. | 64.6 (NA) — Only 1 participant evaluable.
  AR00426032, C1 D1: 4 hrs: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 23 | 1 | 0
  AR00426032, C1 D1: 4 hrs |  |  |  |  |  |  | 9.40 (NA) — Only 1 participant evaluable. | 4.09 (NA) — Only 1 participant evaluable. | 6.71 (145.3) |  | 12.3 (75.3) | 4.61 (NA) — Only 1 participant evaluable. |
  AR00426032, C1 D8: Pre-dose: number analyzed (Participants) | 3 | 2 | 1 | 3 | 0 | 4 | 1 | 1 | 2 | 1 | 21 | 1 | 0
  AR00426032, C1 D8: Pre-dose | 3.98 (31.9) | 2.95 (165.3) | 1.21 (NA) — Only 1 participant evaluable. | 7.10 (122.1) |  | 6.34 (54.5) | 6.15 (NA) — Only 1 participant evaluable. | 1.10 (NA) — Only 1 participant evaluable. | 1.73 (48.7) | 2.09 (NA) — Only 1 participant evaluable. | 5.50 (62.6) | 2.14 (NA) — Only 1 participant evaluable. |
  AR00426032, C1 D15: Pre-dose: number analyzed (Participants) | 3 | 2 | 1 | 4 | 1 | 4 | 1 | 1 | 2 | 0 | 22 | 1 | 0
  AR00426032, C1 D15: Pre-dose | 3.14 (74.5) | 3.80 (111.9) | 1.21 (NA) — Only 1 participant evaluable. | 11.5 (39.5) | 4.36 (NA) — Only 1 participant evaluable. | 5.45 (42.2) | 4.16 (NA) — Only 1 participant evaluable. | NA (NA) — Only 1 participant evaluable. | 3.81 (NA) — Out of 2, 1 participant had BLQ value. |  | 4.19 (79.2) | 1.09 (NA) — Only 1 participant evaluable. |
  AR00426032, C1 D15: 0.5 hr: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 0 | 22 | 0 | 0
  AR00426032, C1 D15: 0.5 hr | 6.66 (43.2) | 7.43 (455.1) | 8.21 (NA) — Only 1 participant evaluable. | 13.1 (97.8) | 11.4 (NA) — Only 1 participant evaluable. | 9.80 (75.7) | 7.31 (NA) — Only 1 participant evaluable. | 4.35 (NA) — Only 1 participant evaluable. | 6.16 (490.6) |  | 7.81 (119.0) |  |
  AR00426032, C1 D15: 1.5 hrs: number analyzed (Participants) | 3 | 2 | 1 | 5 | 0 | 4 | 1 | 1 | 2 | 0 | 22 | 0 | 0
  AR00426032, C1 D15: 1.5 hrs | 24.9 (92.2) | 13.2 (1550.1) | 15.8 (NA) — Only 1 participant evaluable. | 27.9 (85.6) |  | 41.1 (25.7) | 12.9 (NA) — Only 1 participant evaluable. | 12.6 (NA) — Only 1 participant evaluable. | 16.1 (151.9) |  | 18.3 (135.9) |  |
  AR00426032, C1 D15: 2.5 hrs: number analyzed (Participants) | 3 | 2 | 1 | 5 | 0 | 4 | 1 | 1 | 1 | 0 | 22 | 1 | 0
  AR00426032, C1 D15: 2.5 hrs | 18.5 (77.0) | 11.3 (447.2) | 7.75 (NA) — Only 1 participant evaluable. | 18.5 (88.4) |  | 34.3 (51.3) | 9.71 (NA) — Only 1 participant evaluable. | 8.51 (NA) — Only 1 participant evaluable. | 16.2 (NA) — Only 1 participant evaluable. |  | 18.5 (81.2) | 4.73 (NA) — Only 1 participant evaluable. |
  AR00426032, C1 D15: 4 hrs: number analyzed (Participants) | 3 | 2 | 1 | 4 | 1 | 4 | 1 | 0 | 2 | 0 | 23 | 0 | 0
  AR00426032, C1 D15: 4 hrs | 11.8 (40.3) | 9.98 (142.4) | 3.15 (NA) — Only 1 participant evaluable. | 9.46 (142.7) | 22.6 (NA) — Only 1 participant evaluable. | 19.3 (76.9) | 6.76 (NA) — Only 1 participant evaluable. |  | 5.21 (81.9) |  | 12.2 (78.7) |  |
  AR00426032, C1 D15: 6 hrs: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 0 | 20 | 0 | 0
  AR00426032, C1 D15: 6 hrs | 6.86 (61.8) | 7.66 (117.7) | 1.82 (NA) — Only 1 participant evaluable. | 6.90 (142.3) | 8.89 (NA) — Only 1 participant evaluable. | 9.66 (71.5) | 5.82 (NA) — Only 1 participant evaluable. | 2.52 (NA) — Only 1 participant evaluable. | 3.07 (95.0) |  | 7.41 (80.2) |  |
  AR00426032b, C1 D15: 8 hrs: number analyzed (Participants) | 3 | 2 | 0 | 5 | 1 | 3 | 1 | 1 | 2 | 0 | 20 | 0 | 0
  AR00426032b, C1 D15: 8 hrs | 5.94 (76.7) | 5.24 (70.7) |  | 6.49 (124.9) | 8.06 (NA) — Only 1 participant evaluable. | 8.87 (76.5) | 5.12 (NA) — Only 1 participant evaluable. | 1.95 (NA) — Only 1 participant evaluable. | 2.67 (72.9) |  | 6.73 (75.0) |  |
  AR00426032, C1 D16: 24 hrs: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 0 | 22 | 1 | 0
  AR00426032, C1 D16: 24 hrs | 3.99 (61.8) | 2.92 (159.3) | 1.27 (NA) — Only 1 participant evaluable. | 7.79 (87.5) | 1.44 (NA) — Only 1 participant evaluable. | 4.75 (25.4) | 6.53 (NA) — Only 1 participant evaluable. | 1.08 (NA) — Only 1 participant evaluable. | 3.19 (NA) — Only 1 participant evaluable. |  | 4.70 (80.2) | 1.56 (NA) — Only 1 participant evaluable. |
  AR00426032, C1 D21: Pre-dose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 17 | 1 | 1
  AR00426032, C1 D21: Pre-dose |  |  | NA (NA) — Participant had BLQ value. |  |  |  | 3.66 (NA) — Only 1 participant evaluable. | 1.47 (NA) — Only 1 participant evaluable. | 3.18 (NA) — Out of 2, 1 participant had BLQ value. | 1.13 (NA) — Only 1 participant evaluable. | 6.64 (56.1) | 1.65 (NA) — Only 1 participant evaluable. | 3.11 (NA) — Only 1 participant evaluable.
  AR00426032, C2 D1: Pre-dose: number analyzed (Participants) | 3 | 2 | 1 | 5 | 0 | 3 | 1 | 1 | 2 | 1 | 15 | 1 | 1
  AR00426032, C2 D1: Pre-dose | 6.23 (82.0) | 3.51 (36.8) | NA (NA) — Participant had BLQ value. | 13.5 (116.8) |  | 5.71 (44.2) | 4.32 (NA) — Only 1 participant evaluable. | 2.06 (NA) — Only 1 participant evaluable. | 4.09 (NA) — Out of 2, 1 participant had BLQ value. | 3.99 (NA) — Only 1 participant evaluable. | 4.03 (58.1) | NA (NA) — Participant had below BLQ value. | 17.8 (NA) — Only 1 participant evaluable.
  AR00426032, C2 D15: Pre-dose: number analyzed (Participants) | 1 | 1 | 1 | 4 | 1 | 4 | 1 | 1 | 2 | 1 | 14 | 1 | 1
  AR00426032, C2 D15: Pre-dose | 9.97 (NA) — Only 1 participant evaluable. | 7.52 (NA) — Only 1 participant evaluable. | 1.07 (NA) — Only 1 participant evaluable. | 3.27 (65.1) | 1.74 (NA) — Only 1 participant evaluable. | 4.23 (62.5) | 8.54 (NA) — Only 1 participant evaluable. | 1.63 (NA) — Only 1 participant evaluable. | 1.99 (NA) — Only 1 participant evaluable. | 1.19 (NA) — Only 1 participant evaluable. | 5.69 (57.0) | 1.33 (NA) — Only 1 participant evaluable. | 3.74 (NA) — Only 1 participant evaluable.
  AR00426032 C3 D1: Pre-dose: number analyzed (Participants) | 1 | 0 | 1 | 2 | 0 | 4 | 1 | 1 | 0 | 0 | 15 | 1 | 0
  AR00426032 C3 D1: Pre-dose | 9.74 (NA) — Only 1 participant evaluable. |  | NA (NA) — Participant had BLQ value. | 6.15 (NA) — Out of 2, 1 participant had BLQ value. |  | 4.35 (42.3) | 4.50 (NA) — Only 1 participant evaluable. | 1.09 (NA) — Only 1 participant evaluable. |  |  | 4.46 (70.2) | 1.73 (NA) — Only 1 participant evaluable. |
  AR00426032, C4 D1: Pre-dose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 4 | 0 | 0
  AR00426032, C4 D1: Pre-dose | 7.10 (NA) — Only 1 participant evaluable. |  |  |  |  | 5.70 (11.8) | 5.43 (NA) — Only 1 participant evaluable. | 2.78 (NA) — Only 1 participant evaluable. |  |  | 5.78 (83.0) |  |
  AR00426032, C5 D1: Pre-dose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 5 | 0 | 0
  AR00426032, C5 D1: Pre-dose | 6.05 (NA) — Only 1 participant evaluable. |  |  |  |  |  | 8.89 (NA) — Only 1 participant evaluable. | 1.36 (NA) — Only 1 participant evaluable. |  |  | 6.11 (67.8) |  |
  AR00426032, EOT: number analyzed (Participants) | 2 | 1 | 1 | 3 | 1 | 4 | 1 | 1 | 2 | 1 | 20 | 0 | 0
  AR00426032, EOT | NA (NA) — All participants had BLQ value. | NA (NA) — Participant had BLQ value. | NA (NA) — Participant had BLQ value. | NA (NA) — All participants had BLQ value. | NA (NA) — Participant had BLQ value. | 6.68 (80.1) | 3.77 (NA) — Only 1 participant evaluable. | 1.48 (NA) — Only 1 participant evaluable. | 3.65 (NA) — Out of 2, 1 participant had BLQ value. | NA (NA) — Participant had BLQ value. | 4.24 (85.5) |  |

33. Secondary Outcome: Plasma Concentration for Ribociclib (LEE) and Its Metabolite: Part II
Description: LEQ803 is metabolite of ribociclib. Maximum treatment exposure for Part II was of 97.0 weeks.
Time Frame: as for outcome 30
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part II: Encorafenib 100 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 600 mg | Part II: Encorafenib 300 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Ribociclib 600 mg
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 29 | 1 | 1
Nanogram per milliliter
  Ribociclib, C1 D1: 1.5 hrs: number analyzed (Participants) | 1 | 1 | 2 | 0 | 21 | 1 | 1
  Ribociclib, C1 D1: 1.5 hrs | 220 (NA) — Only 1 participant evaluable. | 117 (NA) — Only 1 participant evaluable. | 107 (40.6) |  | 230 (119.7) | 185 (NA) — Only 1 participant evaluable. | 784 (NA) — Only 1 participant evaluable.
  Ribociclib, C1 D1: 4 hrs: number analyzed (Participants) | 1 | 1 | 3 | 0 | 24 | 1 | 0
  Ribociclib, C1 D1: 4 hrs | 213 (NA) — Only 1 participant evaluable. | 84.5 (NA) — Only 1 participant evaluable. | 205 (96.0) |  | 354 (58.5) | 268 (NA) — Only 1 participant evaluable. |
  Ribociclib, C1 D8: Pre-dose: number analyzed (Participants) | 1 | 1 | 2 | 0 | 22 | 1 | 1
  Ribociclib, C1 D8: Pre-dose | 77.4 (NA) — Only 1 participant evaluable. | 32.3 (NA) — Only 1 participant evaluable. | 30.7 (33.5) |  | 100 (49.9) | 80.5 (NA) — Only 1 participant evaluable. | 127 (NA) — Only 1 participant evaluable.
  Ribociclib, C1 D15: Pre-dose: number analyzed (Participants) | 1 | 1 | 2 | 0 | 25 | 1 | 0
  Ribociclib, C1 D15: Pre-dose | 98.4 (NA) — Only 1 participant evaluable. | 28.2 (NA) — Only 1 participant evaluable. | 30.7 (24.9) |  | 104 (54.2) | 64.7 |
  Ribociclib, C1 D15: 0.5 hr: number analyzed (Participants) | 1 | 1 | 2 | 0 | 24 | 0 | 0
  Ribociclib, C1 D15: 0.5 hr | 86.1 (NA) — Only 1 participant evaluable. | 59.7 (NA) — Only 1 participant evaluable. | 35.4 (66.6) |  | 179 (65.0) |  |
  Ribociclib, C1 D15: 1.5 hrs: number analyzed (Participants) | 1 | 1 | 2 | 0 | 24 | 0 | 0
  Ribociclib, C1 D15: 1.5 hrs | 204 (NA) — Only 1 participant evaluable. | 95.9 (NA) — Only 1 participant evaluable. | 200 (240.3) |  | 508 (95.2) |  |
  Ribociclib, C1 D15: 2.5 hrs: number analyzed (Participants) | 1 | 1 | 1 | 0 | 24 | 1 | 0
  Ribociclib, C1 D15: 2.5 hrs | 321 (NA) — Only 1 participant evaluable. | 126 (NA) — Only 1 participant evaluable. | 718 (NA) — Only 1 participant evaluable. |  | 627 (68.3) | 393 (NA) — Only 1 participant evaluable. |
  Ribociclib, C1 D15: 4 hrs: number analyzed (Participants) | 1 | 0 | 2 | 0 | 25 | 0 | 0
  Ribociclib, C1 D15: 4 hrs | 368 (NA) — Only 1 participant evaluable. |  | 341 (42.9) |  | 707 (62.2) |  |
  Ribociclib, C1 D15: 6 hrs: number analyzed (Participants) | 1 | 1 | 2 | 0 | 23 | 0 | 0
  Ribociclib, C1 D15: 6 hrs | 434 (NA) — Only 1 participant evaluable. | 109 (NA) — Only 1 participant evaluable. | 239 (37.2) |  | 578 (55.9) |  |
  Ribociclib, C1 D15: 8 hrs: number analyzed (Participants) | 1 | 1 | 2 | 0 | 21 | 0 | 0
  Ribociclib, C1 D15: 8 hrs | 311 (NA) — Only 1 participant evaluable. | 83.6 (NA) — Only 1 participant evaluable. | 182 (27.1) |  | 477 (55.2) |  |
  Ribociclib, C1 D16: 24 hrs: number analyzed (Participants) | 1 | 1 | 2 | 0 | 24 | 1 | 0
  Ribociclib, C1 D16: 24 hrs | 94.0 (NA) — Only 1 participant evaluable. | 25.6 (NA) — Only 1 participant evaluable. | 52.7 (90.4) |  | 120 (64.9) | 91.8 (NA) — Only 1 participant evaluable. |
  Ribociclib, C1 D21: Pre-dose: number analyzed (Participants) | 1 | 0 | 1 | 0 | 10 | 1 | 1
  Ribociclib, C1 D21: Pre-dose | 105 (NA) — Only 1 participant evaluable. |  | 102 (NA) — Only 1 participant evaluable. |  | 112 (75.8) | 69.9 (NA) — Only 1 participant evaluable. | 115 (NA) — Only 1 participant evaluable.
  Ribociclib, C2 D1: Pre-dose: number analyzed (Participants) | 1 | 1 | 1 | 1 | 16 | 0 | 1
  Ribociclib, C2 D1: Pre-dose | NA (NA) — Participant had BLQ value. | 19.5 (NA) — Only 1 participant evaluable. | 1.59 (NA) — Only 1 participant evaluable. | 1.07 (NA) — Only 1 participant evaluable. | 7.00 (377.8) |  | 132 (NA) — Only 1 participant evaluable.
  Ribociclib, C2 D15: Pre-dose: number analyzed (Participants) | 1 | 1 | 2 | 1 | 15 | 1 | 1
  Ribociclib, C2 D15: Pre-dose | 103 (NA) — Only 1 participant evaluable. | 41.5 (NA) — Only 1 participant evaluable. | 53.7 (51.2) | 36.0 (NA) — Only 1 participant evaluable. | 107 (59.4) | 113 (NA) — Only 1 participant evaluable. | 102 (NA) — Only 1 participant evaluable.
  Ribociclib, C3 D1: Pre-dose: number analyzed (Participants) | 1 | 1 | 0 | 0 | 11 | 0 | 0
  Ribociclib, C3 D1: Pre-dose | 1.16 (NA) — Only 1 participant evaluable. | NA (NA) — Participant had BLQ value. |  |  | 4.06 (172.4) |  |
  Ribociclib, C4 D1: Pre-dose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 2 | 0 | 0
  Ribociclib, C4 D1: Pre-dose | 1.22 (NA) — Only 1 participant evaluable. |  |  |  | 1.59 (31.6) |  |
  Ribociclib, C5 D1: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Ribociclib, C5 D1: Pre-dose |  |  |  |  | 2.16 (35.5) |  |
  Ribociclib, EOT: number analyzed (Participants) | 1 | 1 | 2 | 1 | 21 | 0 | 1
  Ribociclib, EOT | 1.94 (NA) — Only 1 participant evaluable. | 60.3 (NA) — Only 1 participant evaluable. | 1.49 (NA) — One participant had BLQ value. | 45.8 (NA) — Only 1 participant evaluable. | 29.0 (292.1) |  | 22.8 (NA) — Only 1 participant evaluable.
  LEQ803, C1 D1: 1.5 hrs: number analyzed (Participants) | 1 | 1 | 2 | 0 | 21 | 1 | 1
  LEQ803, C1 D1: 1.5 hrs | 57.1 (NA) — Only 1 participant evaluable. | 70.2 (NA) — Only 1 participant evaluable. | 68.2 (2.4) |  | 47.5 (97.4) | 59.0 (NA) — Only 1 participant evaluable. | 63.6 (NA) — Only 1 participant evaluable.
  LEQ803, C1 D1: 4 hrs: number analyzed (Participants) | 1 | 1 | 3 | 0 | 24 | 1 | 0
  LEQ803, C1 D1: 4 hrs | 65.2 (NA) — Only 1 participant evaluable. | 50.8 (NA) — Only 1 participant evaluable. | 73.5 (20.4) |  | 81.1 (55.6) | 63.2 (NA) — Only 1 participant evaluable. |
  LEQ803, C1 D8: Pre-dose: number analyzed (Participants) | 1 | 1 | 2 | 0 | 22 | 1 | 1
  LEQ803, C1 D8: Pre-dose | 64.3 (NA) — Only 1 participant evaluable. | 49.3 (NA) — Only 1 participant evaluable. | 38.1 (9.1) |  | 53.7 (36.5) | 47.2 | 71.2
  LEQ803, C1 D15: Pre-dose: number analyzed (Participants) | 1 | 1 | 2 | 0 | 25 | 1 | 0
  LEQ803, C1 D15: Pre-dose | 76.0 (NA) — Only 1 participant evaluable. | 37.1 (NA) — Only 1 participant evaluable. | 32.9 (25.7) |  | 55.1 (33.9) | 49.2 (NA) — Only 1 participant evaluable. |
  LEQ803, C1 D15: 0.5 hr: number analyzed (Participants) | 1 | 1 | 2 | 0 | 24 | 0 | 0
  LEQ803, C1 D15: 0.5 hr | 75.5 (NA) — Only 1 participant evaluable. | 39.5 (NA) — Only 1 participant evaluable. | 32.1 (0.7) |  | 60.8 (36.9) |  |
  LEQ803, C1 D15: 1.5 hrs: number analyzed (Participants) | 1 | 1 | 2 | 0 | 24 | 0 | 0
  LEQ803, C1 D15: 1.5 hrs | 92.3 (NA) — Only 1 participant evaluable. | 72.6 (NA) — Only 1 participant evaluable. | 82.7 (0.7) |  | 112 (46.9) |  |
  LEQ803, C1 D15: 2.5 hrs: number analyzed (Participants) | 1 | 1 | 1 | 0 | 24 | 1 | 0
  LEQ803, C1 D15: 2.5 hrs | 130 (NA) — Only 1 participant evaluable. | 92.5 (NA) — Only 1 participant evaluable. | 126 (NA) — Only 1 participant evaluable. |  | 133 (45.4) | 137 (NA) — Only 1 participant evaluable. |
  LEQ803, C1 D15: 4 hrs: number analyzed (Participants) | 1 | 0 | 2 | 0 | 25 | 0 | 0
  LEQ803, C1 D15: 4 hrs | 138 (NA) — Only 1 participant evaluable. |  | 140 (23.4) |  | 152 (31.2) |  |
  LEQ803, C1 D15: 6 hrs: number analyzed (Participants) | 1 | 1 | 2 | 0 | 23 | 0 | 0
  LEQ803, C1 D15: 6 hrs | 175 (NA) — Only 1 participant evaluable. | 90.2 (NA) — Only 1 participant evaluable. | 111 (27.6) |  | 145 (27.2) |  |
  LEQ803, C1 D15: 8 hrs: number analyzed (Participants) | 1 | 1 | 2 | 0 | 21 | 0 | 0
  LEQ803, C1 D15: 8 hrs | 135 (NA) — Only 1 participant evaluable. | 79.8 (NA) — Only 1 participant evaluable. | 95.2 (50.1) |  | 128 (27.6) |  |
  LEQ803, C1 D16: 24 hrs: number analyzed (Participants) | 1 | 1 | 2 | 0 | 24 | 1 | 0
  LEQ803, C1 D16: 24 hrs | 84.5 (NA) — Only 1 participant evaluable. | 46.8 (NA) — Only 1 participant evaluable. | 42.5 (13.8) |  | 63.1 (36.1) | 59.6 (NA) — Only 1 participant evaluable. |
  LEQ803, C1 D21: Pre-dose: number analyzed (Participants) | 1 | 0 | 1 | 0 | 10 | 1 | 1
  LEQ803, C1 D21: Pre-dose | 73.8 (NA) — Only 1 participant evaluable. |  | 43.7 (NA) — Only 1 participant evaluable. |  | 58.1 (39.1) | 52.9 (NA) — Only 1 participant evaluable. | 80.2 (NA) — Only 1 participant evaluable.
  LEQ803, C2 D1: Pre-dose: number analyzed (Participants) | 1 | 1 | 1 | 1 | 16 | 0 | 1
  LEQ803, C2 D1: Pre-dose | 6.68 (NA) — Only 1 participant evaluable. | 14.5 (NA) — Only 1 participant evaluable. | 4.10 (NA) — Only 1 participant evaluable. | 2.70 (NA) — Only 1 participant evaluable. | 8.48 (154.5) |  | 80.8 (NA) — Only 1 participant evaluable.
  LEQ803, C2 D15: Pre-dose: number analyzed (Participants) | 1 | 1 | 2 | 1 | 15 | 1 | 1
  LEQ803, C2 D15: Pre-dose | 90.0 (NA) — Only 1 participant evaluable. | 45.6 (NA) — Only 1 participant evaluable. | 45.7 (6.8) | 28.0 (NA) — Only 1 participant evaluable. | 58.3 (42.7) | 66.8 (NA) — Only 1 participant evaluable. | 61.1 (NA) — Only 1 participant evaluable.
  LEQ803, C3 D1: Pre-dose: number analyzed (Participants) | 1 | 1 | 0 | 0 | 11 | 0 | 0
  LEQ803, C3 D1: Pre-dose | 7.88 (NA) — Only 1 participant evaluable. | 2.75 (NA) — Only 1 participant evaluable. |  |  | 7.57 (61.4) |  |
  LEQ803, C4 D1: Pre-dose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 2 | 0 | 0
  LEQ803, C4 D1: Pre-dose | 7.19 (NA) — Only 1 participant evaluable. |  |  |  | 5.72 (6.9) |  |
  LEQ803, C5 D1: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 0
  LEQ803, C5 D1: Pre-dose |  |  |  |  | 6.07 (28.9) |  |
  LEQ803, EOT: number analyzed (Participants) | 1 | 1 | 2 | 1 | 21 | 0 | 1
  LEQ803, EOT | 10.4 (NA) — Only 1 participant evaluable. | 69.3 (NA) — Only 1 participant evaluable. | 5.06 (4.6) | 23.5 (NA) — Only 1 participant evaluable. | 20.6 (152.2) |  | 31.2 (NA) — Only 1 participant evaluable.

34. Secondary Outcome: Plasma Concentration for Infigratinib (BGJ) and Its Metabolites: Part II
Description: BHS697 and CQM157 are metabolites of infigratinib. Maximum treatment exposure for Part II was of 97.0 weeks.
Time Frame: C1 (1.5 hrs post-dose on D1; pre-dose on D8; pre-dose, 0.5, 1.5, 2.5, 4, 6 hrs post-dose on D15; 24 hrs post-dose on D16; pre-dose on D21); C2 (pre-dose on D1 and D15); C3 pre-dose on D1; EOT
Population: PAS consisted of all participants who had at least one blood sample providing evaluable PK data. Here, "Number Analyzed" signifies number of participants evaluable for specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Infigratinib 75 mg
Number analyzed (Participants) | 1
Nanogram per milliliter
  Infigratinib, C1 D1: 1.5 hrs | 15.0 (NA) — Only 1 participant evaluable.
  Infigratinib, C1 D8: Pre-dose | 2.67 (NA) — Only 1 participant evaluable.
  Infigratinib, C1 D15: Pre-dose | 2.49 (NA) — Only 1 participant evaluable.
  Infigratinib, C1 D15: 0.5 hr | 3.39 (NA) — Only 1 participant evaluable.
  Infigratinib, C1 D15: 1.5 hrs | 15.2 (NA) — Only 1 participant evaluable.
  Infigratinib, C1 D15: 2.5 hrs | 27.5 (NA) — Only 1 participant evaluable.
  Infigratinib, C1 D15: 4 hrs | 24.7 (NA) — Only 1 participant evaluable.
  Infigratinib, C1 D15: 6 hrs | 20.5 (NA) — Only 1 participant evaluable.
  Infigratinib, C1 D16: 24 hrs: number analyzed (Participants) | 0
  Infigratinib, C1 D21: Pre-dose | 2.05 (NA) — Only 1 participant evaluable.
  Infigratinib, C2 D1: Pre-dose | NA (NA) — Participant had BLQ value.
  Infigratinib, C2 D15: Pre-dose | 4.65 (NA) — Only 1 participant evaluable.
  Infigratinib, C3 D1: Pre-dose | NA (NA) — Participant had BLQ value.
  Infigratinib, EOT | 2.42 (NA) — Only 1 participant evaluable.
  BHS697, C1 D1: 1.5 hrs | 4.83 (NA) — Only 1 participant evaluable.
  BHS697, C1 D8: Pre-dose | 2.17 (NA) — Only 1 participant evaluable.
  BHS697, C1 D15: Pre-dose | 1.64 (NA) — Only 1 participant evaluable.
  BHS697, C1 D15: 0.5 hr | 2.14 (NA) — Only 1 participant evaluable.
  BHS697, C1 D15: 1.5 hrs | 6.83 (NA) — Only 1 participant evaluable.
  BHS697, C1 D15: 2.5 hrs | 8.53 (NA) — Only 1 participant evaluable.
  BHS697, C1 D15: 4 hrs | 6.89 (NA) — Only 1 participant evaluable.
  BHS697, C1 D15: 6 hrs | 5.57 (NA) — Only 1 participant evaluable.
  BHS697, C1 D16: 24 hrs: number analyzed (Participants) | 0
  BHS697, C1 D21: Pre-dose | 1.37 (NA) — Only 1 participant evaluable.
  BHS697, C2 D1: Pre-dose | NA (NA) — Participant had BLQ value.
  BHS697, C2 D15: Pre-dose | 2.83 (NA) — Only 1 participant evaluable.
  BHS697, C3 D1: Pre-dose | NA (NA) — Participant had BLQ value.
  BHS697, EOT | 1.69 (NA) — Only 1 participant evaluable.
  CQM157, C1 D1: 1.5 hrs | 13.0 (NA) — Only 1 participant evaluable.
  CQM157, C1 D8: Pre-dose | 14.1 (NA) — Only 1 participant evaluable.
  CQM157, C1 D15: Pre-dose | 11.1 (NA) — Only 1 participant evaluable.
  CQM157, C1 D15: 0.5 hr | 12.0 (NA) — Only 1 participant evaluable.
  CQM157, C1 D15: 1.5 hrs | 21.3 (NA) — Only 1 participant evaluable.
  CQM157, C1 D15: 2.5 hrs | 28.3 (NA) — Only 1 participant evaluable.
  CQM157, C1 D15: 4 hrs | 25.0 (NA) — Only 1 participant evaluable.
  CQM157, C1 D15: 6 hrs | 32.2 (NA) — Only 1 participant evaluable.
  CQM157, C1 D16: 24 hrs: number analyzed (Participants) | 0
  CQM157, C1 D21: Pre-dose | 9.65 (NA) — Only 1 participant evaluable.
  CQM157, C2 D1: Pre-dose | NA (NA) — Participant had BLQ value.
  CQM157, C2 D15: Pre-dose | 15.5 (NA) — Only 1 participant evaluable.
  CQM157, C3 D1: Pre-dose | NA (NA) — Participant had BLQ value.
  CQM157, EOT | 11.9 (NA) — Only 1 participant evaluable.

35. Secondary Outcome: Plasma Concentration for Capmatinib (INC): Part II
Description: Maximum treatment exposure for Part II was of 97.0 weeks.
Time Frame: C1 (1.5 hrs post-dose on D1; pre-dose on D8; pre-dose, 0.5, 1.5, 2.5, 4, 6, 8 hrs post-dose on D15; 24 hrs post-dose on D16); C2 (pre-dose on D1 and D15); C3 pre-dose on D1; C4 pre-dose on D1; C5 pre-dose on D1; EOT
Population: PAS consisted of all participants who had at least one blood sample providing evaluable PK data. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable for specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 200 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 300 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 400 mg
Number analyzed (Participants) | 5 | 1 | 5
Nanogram per milliliter
  C1 D1: 1.5 hrs: number analyzed (Participants) | 3 | 1 | 2
  C1 D1: 1.5 hrs | 362 (268.6) | 3600 (NA) — Only 1 participant evaluable. | 715 (133.2)
  C1 D8: Pre-dose: number analyzed (Participants) | 3 | 1 | 4
  C1 D8: Pre-dose | 74.3 (97.2) | 44.4 (NA) — Only 1 participant evaluable. | 129 (49.4)
  C1 D15: Pre-dose: number analyzed (Participants) | 4 | 1 | 4
  C1 D15: Pre-dose | 89.3 (35.7) | 71.4 (NA) — Only 1 participant evaluable. | 173 (41.2)
  C1 D15: 0.5 hr: number analyzed (Participants) | 5 | 1 | 4
  C1 D15: 0.5 hr | 196 (103.8) | 1880 (NA) — Only 1 participant evaluable. | 314 (49.0)
  C1 D15: 1.5 hrs: number analyzed (Participants) | 5 | 1 | 4
  C1 D15: 1.5 hrs | 636 (78.2) | 3670 (NA) — Only 1 participant evaluable. | 1830 (38.3)
  C1 D15: 2.5 hrs: number analyzed (Participants) | 5 | 0 | 4
  C1 D15: 2.5 hrs | 545 (81.2) |  | 1530 (18.4)
  C1 D15: 4 hrs: number analyzed (Participants) | 4 | 1 | 4
  C1 D15: 4 hrs | 401 (17.3) | 1230 (NA) — Only 1 participant evaluable. | 950 (39.1)
  C1 D15: 6 hrs: number analyzed (Participants) | 5 | 1 | 4
  C1 D15: 6 hrs | 157 (63.2) | 264 (NA) — Only 1 participant evaluable. | 487 (23.3)
  C1 D15: 8 hrs: number analyzed (Participants) | 5 | 1 | 3
  C1 D15: 8 hrs | 120 (50.0) | 268 (NA) — Only 1 participant evaluable. | 390 (10.5)
  C1 D16: 24 hrs: number analyzed (Participants) | 5 | 1 | 4
  C1 D16: 24 hrs | 79.6 (103.1) | 58.1 (NA) — Only 1 participant evaluable. | 269 (68.7)
  C2 D1: Pre-dose: number analyzed (Participants) | 5 | 1 | 3
  C2 D1: Pre-dose | 151 (107.6) | 38.7 (NA) — Only 1 participant evaluable. | 227 (42.0)
  C2 D15: Pre-dose: number analyzed (Participants) | 3 | 1 | 3
  C2 D15: Pre-dose | 65.2 (31.0) | 50.5 (NA) — Only 1 participant evaluable. | 166 (80.9)
  C3 D1: Pre-dose: number analyzed (Participants) | 2 | 0 | 3
  C3 D1: Pre-dose | 114 (113.4) |  | 96.5 (17.9)
  C4 D1: Pre-dose: number analyzed (Participants) | 0 | 0 | 3
  C4 D1: Pre-dose |  |  | 175 (44.8)
  C5 D1: Pre-dose: number analyzed (Participants) | 0 | 1 | 0
  C5 D1: Pre-dose |  | 41.8 (NA) — Only 1 participant evaluable. |
  EOT: number analyzed (Participants) | 3 | 1 | 4
  EOT | NA (NA) — All participants had BLQ values. | NA (NA) — Participant had BLQ value. | 65.4 (155.0)

36. Secondary Outcome: Plasma Concentration for Buparlisib (BKM): Part II
Description: Maximum treatment exposure for Part II was of 97.0 weeks.
Time Frame: as for outcome 35
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 60 mg: Participants received encorafenib 450 mg QD and binimetinib 45 mg BID and buparlisib 60 mg QD.
Arm/Group | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 60 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 90 mg
Number analyzed (Participants) | 3 | 3
Nanogram per milliliter
  C1 D1: 1.5 hrs: number analyzed (Participants) | 1 | 1
  C1 D1: 1.5 hrs | 213 (NA) — Only 1 participant evaluable. | 213 (NA) — Only 1 participant evaluable.
  C1 D8: Pre-dose: number analyzed (Participants) | 3 | 2
  C1 D8: Pre-dose | 45.0 (75.2) | 119 (3.6)
  C1 D15: Pre-dose: number analyzed (Participants) | 3 | 2
  C1 D15: Pre-dose | 49.7 (115.9) | 97.3 (16.2)
  C1 D15: 0.5 hr: number analyzed (Participants) | 3 | 2
  C1 D15: 0.5 hr | 139 (13.4) | 229 (21.5)
  C1 D15: 1.5 hrs: number analyzed (Participants) | 3 | 2
  C1 D15: 1.5 hrs | 266 (51.5) | 312 (10.9)
  C1 D15: 2.5 hrs: number analyzed (Participants) | 3 | 2
  C1 D15: 2.5 hrs | 176 (42.2) | 268 (11.9)
  C1 D15: 4 hrs: number analyzed (Participants) | 3 | 2
  C1 D15: 4 hrs | 115 (44.0) | 235 (39.4)
  C1 D15: 6 hrs: number analyzed (Participants) | 3 | 2
  C1 D15: 6 hrs | 94.2 (40.0) | 171 (26.4)
  C1 D15: 8 hrs: number analyzed (Participants) | 3 | 2
  C1 D15: 8 hrs | 87.4 (63.9) | 111 (25.5)
  C1 D16: 24 hrs: number analyzed (Participants) | 3 | 2
  C1 D16: 24 hrs | 41.8 (82.9) | 101 (1.4)
  C2 D1: Pre-dose: number analyzed (Participants) | 3 | 2
  C2 D1: Pre-dose | 54.7 (134.9) | 110 (51.2)
  C2 D15: Pre-dose: number analyzed (Participants) | 1 | 1
  C2 D15: Pre-dose | 99.3 (NA) — Only 1 participant evaluable. | 138 (NA) — Only 1 participant evaluable.
  C3 D1: Pre-dose: number analyzed (Participants) | 1 | 0
  C3 D1: Pre-dose | 81.2 (NA) — Only 1 participant evaluable. |
  C4 D1: Pre-dose: number analyzed (Participants) | 1 | 0
  C4 D1: Pre-dose | 73.2 (NA) — Only 1 participant evaluable. |
  C5 D1: Pre-dose: number analyzed (Participants) | 1 | 0
  C5 D1: Pre-dose | 122 (NA) — Only 1 participant evaluable. |
  EOT: number analyzed (Participants) | 2 | 1
  EOT | 1.84 (53.4) | NA (NA) — Participant had BLQ value.

37. Secondary Outcome: Maximum Observed Plasma Concentration at Steady State (Cmax,ss) for Encorafenib, Binimetinib, Binimetinib Metabolite, Ribociclib, Ribociclib Metabolite, Infigratinib, Infigratinib Metabolites, Capmatinib, and Buparlisib: Part II
Time Frame: C1 D15: 0.5 hour ± 10 (minutes) min; 1 hour ± 10 min; 1.5 hour ± 15 min; 2 hour ± 15 min; 2.5 hour ± 15 min; 4 hour ± 30 min; 6 hour ± 30 min; 8 hour ± 60 min; 24 hour ± 2 hour
Population: PAS consisted of all participants who had at least one blood sample providing evaluable PK data. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable for specified study treatment or metabolites for respective arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- Part II: Encorafenib 300 mg/Binimetinib 30 mg + Ribociclib 600 mg: Participants received encorafenib 300 mg QD and binimetinib 30 mg BID and ribociclib 600 mg QD.
Arm/Group | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 60 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 90 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Infigratinib 75 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 200 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 300 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 400 mg | Part II: Encorafenib 100 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 600 mg | Part II: Encorafenib 300 mg/Binimetinib 30 mg + Ribociclib 600 mg
Number analyzed (Participants) | 3 | 3 | 1 | 5 | 1 | 5 | 1 | 1 | 3 | 1 | 29 | 1
Nanogram per milliliter
  Encorafenib: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 1 | 25 | 0
  Encorafenib | 3060 (58.8) | 2150 (54.6) | 2100 (NA) — Only 1 participant evaluable. | 1600 (62.0) | 2890 (NA) — Only 1 participant evaluable. | 2570 (23.0) | 622 (NA) — Only 1 participant evaluable. | 1960 (NA) — Only 1 participant evaluable. | 1860 (32.1) | 2010 (NA) — Only 1 participant evaluable. | 2030 (40.6) |
  Binimetinib: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 1 | 24 | 1
  Binimetinib | 386 (41.1) | 221 (237.6) | 413 (NA) — Only 1 participant evaluable. | 515 (17.0) | 797 (NA) — Only 1 participant evaluable. | 858 (13.0) | 261 (NA) — Only 1 participant evaluable. | 520 (NA) — Only 1 participant evaluable. | 313 (15.9) | 584 (NA) — Only 1 participant evaluable. | 489 (31.3) | 291 (NA) — Only 1 participant evaluable.
  Binimetinib metabolite, AR00426032: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 1 | 24 | 1
  Binimetinib metabolite, AR00426032 | 24.9 (92.2) | 18.1 (591.2) | 15.8 (NA) — Only 1 participant evaluable. | 27.9 (85.6) | 22.6 (NA) — Only 1 participant evaluable. | 47.1 (29.2) | 12.9 (NA) — Only 1 participant evaluable. | 12.6 (NA) — Only 1 participant evaluable. | 16.1 (151.9) | 19.4 (NA) — Only 1 participant evaluable. | 23.7 (94.1) | 9.04 (NA) — Only 1 participant evaluable.
  Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 26 | 1
  Ribociclib |  |  |  |  |  |  | 434 (NA) — Only 1 participant evaluable. | 126 (NA) — Only 1 participant evaluable. | 428 (84.2) | 282 (NA) — Only 1 participant evaluable. | 753 (70.6) | 597 (NA) — Only 1 participant evaluable.
  Ribociclib metabolite, LEQ803: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 26 | 1
  Ribociclib metabolite, LEQ803 |  |  |  |  |  |  | 175 (NA) — Only 1 participant evaluable. | 93.2 (NA) — Only 1 participant evaluable. | 144 (19.2) | 67.5 (NA) — Only 1 participant evaluable. | 156 (36.2) | 138 (NA) — Only 1 participant evaluable.
  Infigratinib: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infigratinib |  |  | 27.5 (NA) — Only 1 participant evaluable. |  |  |  |  |  |  |  |  |
  Infigratinib metabolite, BHS697: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infigratinib metabolite, BHS697 |  |  | 8.53 (NA) — Only 1 participant evaluable. |  |  |  |  |  |  |  |  |
  Infigratinib metabolite, CQM157: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infigratinib metabolite, CQM157 |  |  | 32.2 (NA) — Only 1 participant evaluable. |  |  |  |  |  |  |  |  |
  Capmatinib: number analyzed (Participants) | 0 | 0 | 0 | 5 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
  Capmatinib |  |  |  | 722 (85.3) | 3670 (NA) — Only 1 participant evaluable. | 1920 (31.8) |  |  |  |  |  |
  Buparlisib: number analyzed (Participants) | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Buparlisib | 266 (51.5) | 312 (10.9) |  |  |  |  |  |  |  |  |  |

38. Secondary Outcome: Time to Reach Cmax at Steady State (Tmax, ss) for Encorafenib, Binimetinib, Binimetinib Metabolite, Ribociclib, Ribociclib Metabolite, Infigratinib, Infigratinib Metabolites, Capmatinib, and Buparlisib: Part II
Time Frame: C1 D15: 0.5 hour ± 10 min; 1 hour ± 10 min; 1.5 hour ± 15 min; 2 hour ± 15 min; 2.5 hour ± 15 min; 4 hour ± 30 min; 6 hour ± 30 min; 8 hour ± 60 min; 24 hour ± 2 hour
Population: as for outcome 37
Measure: Median (Full Range); unit: Hour
Arm/Group | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 60 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 90 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Infigratinib 75 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 200 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 300 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 400 mg | Part II: Encorafenib 100 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 600 mg | Part II: Encorafenib 300 mg/Binimetinib 30 mg + Ribociclib 600 mg
Number analyzed (Participants) | 3 | 3 | 1 | 5 | 1 | 5 | 1 | 1 | 3 | 1 | 29 | 1
Hour
  Encorafenib: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 1 | 25 | 0
  Encorafenib | 1.33 [0.58 to 1.50] | 1.54 [1.50 to 1.58] | 1.50 [1.50 to 1.50] | 1.50 [0.50 to 1.53] | 1.50 [1.50 to 1.50] | 1.50 [1.50 to 2.50] | 2.37 [2.37 to 2.37] | 1.47 [1.47 to 1.47] | 1.00 [0.50 to 1.50] | 1.50 [1.50 to 1.50] | 1.58 [0.63 to 6.17] |
  Binimetinib: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 1 | 24 | 1
  Binimetinib | 1.50 [1.33 to 1.67] | 2.75 [1.50 to 4.00] | 1.50 [1.50 to 1.50] | 1.50 [0.50 to 1.58] | 1.50 [1.50 to 1.50] | 1.50 [1.50 to 2.50] | 1.38 [1.38 to 1.38] | 1.47 [1.47 to 1.47] | 1.50 [1.50 to 1.50] | 1.50 [1.50 to 1.50] | 1.58 [0.50 to 4.08] | 1.08 [1.08 to 1.08]
  Binimetinib metabolite, AR00426032: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 1 | 24 | 1
  Binimetinib metabolite, AR00426032 | 1.50 [1.33 to 1.67] | 2.75 [1.50 to 4.00] | 1.50 [1.50 to 1.50] | 1.50 [1.50 to 1.58] | 4.00 [4.00 to 4.00] | 1.92 [1.50 to 2.50] | 1.38 [1.38 to 1.38] | 1.47 [1.47 to 1.47] | 1.50 [1.50 to 1.50] | 1.50 [1.50 to 1.50] | 1.65 [0.67 to 4.08] | 1.08 [1.08 to 1.08]
  Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 26 | 1
  Ribociclib |  |  |  |  |  |  | 5.92 [5.92 to 5.92] | 2.45 [2.45 to 2.45] | 3.18 [2.33 to 4.03] | 1.50 [1.50 to 1.50] | 3.65 [1.50 to 6.00] | 0.50 [0.50 to 0.50]
  Ribociclib metabolite, LEQ803: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 26 | 1
  Ribociclib metabolite, LEQ803 |  |  |  |  |  |  | 5.92 [5.92 to 5.92] | 4.98 [4.98 to 4.98] | 3.18 [2.33 to 4.03] | 1.50 [1.50 to 1.50] | 4.12 [1.55 to 7.00] | 1.08 [1.08 to 1.08]
  Infigratinib: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infigratinib |  |  | 2.50 [2.50 to 2.50] |  |  |  |  |  |  |  |  |
  Infigratinib metabolite, BHS697: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infigratinib metabolite, BHS697 |  |  | 2.50 [2.50 to 2.50] |  |  |  |  |  |  |  |  |
  Infigratinib metabolite, CQM157: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infigratinib metabolite, CQM157 |  |  | 5.75 [5.75 to 5.75] |  |  |  |  |  |  |  |  |
  Capmatinib: number analyzed (Participants) | 0 | 0 | 0 | 5 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
  Capmatinib |  |  |  | 1.53 [1.50 to 2.58] | 1.50 [1.50 to 1.50] | 1.50 [1.50 to 2.50] |  |  |  |  |  |
  Buparlisib: number analyzed (Participants) | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Buparlisib | 1.50 [1.33 to 1.67] | 1.50 [1.50 to 1.50] |  |  |  |  |  |  |  |  |  |

39. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Time Tau at Steady-State (AUCtau,ss) for Encorafenib, Binimetinib, Binimetinib Metabolite, Ribociclib, Ribociclib Metabolite, Capmatinib, and Buparlisib: Part II
Time Frame: as for outcome 38
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 60 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 90 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Infigratinib 75 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 200 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 300 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 400 mg | Part II: Encorafenib 100 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 600 mg | Part II: Encorafenib 300 mg/Binimetinib 30 mg + Ribociclib 600 mg
Number analyzed (Participants) | 3 | 3 | 1 | 5 | 1 | 5 | 1 | 1 | 3 | 1 | 29 | 1
Hour*nanogram per milliliter
  Encorafenib: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 1 | 23 | 0
  Encorafenib | 9080 (42.2) | 10100 (18.4) | 7420 (NA) — Only 1 participant evaluable. | 4990 (42.6) | 10800 (NA) — Only 1 participant evaluable. | 8570 (10.6) | 3490 (NA) — Only 1 participant evaluable. | 6000 (NA) — Only 1 participant evaluable. | 5740 (7.1) | 6200 (NA) — Only 1 participant evaluable. | 11300 (41.1) |
  Binimetinib: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 1 | 23 | 1
  Binimetinib | 1580 (17.0) | 1220 (105.7) | 1260 (NA) — Only 1 participant evaluable. | 2180 (29.4) | 3040 (NA) — Only 1 participant evaluable. | 2760 (4.8) | 1700 (NA) — Only 1 participant evaluable. | 1900 (NA) — Only 1 participant evaluable. | 1140 (21.1) | 1740 (NA) — Only 1 participant evaluable. | 2270 (29.5) | 1470 (NA) — Only 1 participant evaluable.
  Binimetinib metabolite, AR00426032: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 1 | 22 | 1
  Binimetinib metabolite, AR00426032 | 116 (66.8) | 94.4 (222.2) | 42.0 (NA) — Only 1 participant evaluable. | 124 (113.9) | 135 (NA) — Only 1 participant evaluable. | 182 (43.1) | 81.5 (NA) — Only 1 participant evaluable. | 47.0 (NA) — Only 1 participant evaluable. | 57.9 (128.5) | 66.9 (NA) — Only 1 participant evaluable. | 115 (92.6) | 41.1 (NA) — Only 1 participant evaluable.
  Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 22 | 1
  Ribociclib |  |  |  |  |  |  | 5630 (NA) — Only 1 participant evaluable. | 1650 (NA) — Only 1 participant evaluable. | 3730 (62.5) | 2320 (NA) — Only 1 participant evaluable. | 9230 (60.9) | 5960 (NA) — Only 1 participant evaluable.
  Ribociclib metabolite, LEQ803: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 22 | 1
  Ribociclib metabolite, LEQ803 |  |  |  |  |  |  | 2770 (NA) — Only 1 participant evaluable. | 1640 (NA) — Only 1 participant evaluable. | 1900 (24.9) | 930 (NA) — Only 1 participant evaluable. | 2540 (31.3) | 2300 (NA) — Only 1 participant evaluable.
  Capmatinib: number analyzed (Participants) | 0 | 0 | 0 | 5 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
  Capmatinib |  |  |  | 3070 (52.6) | 12200 (NA) — Only 1 participant evaluable. | 8420 (22.0) |  |  |  |  |  |
  Buparlisib: number analyzed (Participants) | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Buparlisib | 2130 (54.6) | 3400 (18.5) |  |  |  |  |  |  |  |  |  |

40. Secondary Outcome: Elimination Half-life at Steady State (t1/2, ss) of Encorafenib, Binimetinib, Binimetinib Metabolite, Ribociclib, Ribociclib Metabolite, Capmatinib, and Buparlisib: Part II
Description: Elimination half-life means the time required for the plasma concentration to decline by 50% during the elimination phase.
Time Frame: as for outcome 38
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 60 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 90 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Infigratinib 75 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 200 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 300 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 400 mg | Part II: Encorafenib 100 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 600 mg | Part II: Encorafenib 300 mg/Binimetinib 30 mg + Ribociclib 600 mg
Number analyzed (Participants) | 3 | 3 | 1 | 5 | 1 | 5 | 1 | 1 | 3 | 1 | 29 | 1
Hour
  Encorafenib: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 1 | 20 | 0
  Encorafenib | 3.75 (0.302) | 5.89 (4.32) | 3.57 (NA) — Only 1 participant evaluable. | 4.18 (1.85) | 3.41 (NA) — Only 1 participant evaluable. | 3.96 (0.233) | 4.27 (NA) — Only 1 participant evaluable. | 3.75 (NA) — Only 1 participant evaluable. | 4.32 (1.62) | 3.83 (NA) — Only 1 participant evaluable. | 3.60 (0.711) |
  Binimetinib: number analyzed (Participants) | 3 | 2 | 1 | 4 | 0 | 4 | 1 | 1 | 2 | 1 | 22 | 0
  Binimetinib | 8.35 (3.52) | 3.48 (0.484) | 1.60 (NA) — Only 1 participant evaluable. | 10.3 (6.29) |  | 5.88 (2.77) | 5.84 (NA) — Only 1 participant evaluable. | 3.82 (NA) — Only 1 participant evaluable. | 5.38 (3.39) | 10.9 (NA) — Only 1 participant evaluable. | 4.13 (1.42) |
  Binimetinib metabolite, AR00426032: number analyzed (Participants) | 3 | 2 | 1 | 2 | 1 | 3 | 0 | 1 | 2 | 0 | 17 | 0
  Binimetinib metabolite, AR00426032 | 6.35 (1.21) | 4.14 (0.683) | 1.59 (NA) — Only 1 participant evaluable. | 7.95 (4.03) | 2.86 (NA) — Only 1 participant evaluable. | 5.64 (2.49) |  | 4.34 (NA) — Only 1 participant evaluable. | 6.24 (4.43) |  | 5.91 (3.00) |
  Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 18 | 1
  Ribociclib |  |  |  |  |  |  |  | 9.01 (NA) — Only 1 participant evaluable. | 8.44 (2.21) | 10.7 (NA) — Only 1 participant evaluable. | 7.77 (1.95) | 10.1 (NA) — Only 1 participant evaluable.
  Ribociclib metabolite, LEQ803: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 11 | 0
  Ribociclib metabolite, LEQ803 |  |  |  |  |  |  |  | 19.9 (NA) — Only 1 participant evaluable. | 14.1 (4.04) | 19.2 (NA) — Only 1 participant evaluable. | 16.0 (4.50) |
  Capmatinib: number analyzed (Participants) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Capmatinib |  |  |  | 2.18 (0.0599) | 2.50 (NA) — Only 1 participant evaluable. | 2.82 (NA) — Only 1 participant evaluable. |  |  |  |  |  |
  Buparlisib: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Buparlisib | 15.4 (4.62) |  |  |  |  |  |  |  |  |  |  |

41. Secondary Outcome: Apparent Total Plasma Clearance at Steady State (Cl, ss/F) of Encorafenib, Binimetinib, Ribociclib, Capmatinib, and Buparlisib: Part II
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: as for outcome 38
Population: PAS consisted of all participants who had at least one blood sample providing evaluable PK data. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable for specified study treatment for respective arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 60 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 90 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Infigratinib 75 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 200 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 300 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 400 mg | Part II: Encorafenib 100 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 600 mg | Part II: Encorafenib 300 mg/ Binimetinib 30 mg + Ribociclib 600 mg
Number analyzed (Participants) | 3 | 3 | 1 | 5 | 1 | 5 | 1 | 1 | 3 | 1 | 29 | 1
Liter per hour
  Encorafenib: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 1 | 20 | 0
  Encorafenib | 49.6 (42.1) | 44.7 (18.4) | 60.7 (NA) — Only 1 participant evaluable. | 40.1 (42.6) | 18.6 (NA) — Only 1 participant evaluable. | 23.4 (10.7) | 28.7 (NA) — Only 1 participant evaluable. | 33.3 (NA) — Only 1 participant evaluable. | 34.9 (6.9) | 32.2 (NA) — Only 1 participant evaluable. | 19.5 (44.3) |
  Binimetinib: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 1 | 23 | 0
  Binimetinib | 28.5 (14.8) | 36.9 (105.7) | 35.6 (NA) — Only 1 participant evaluable. | 20.8 (28.1) | 15.1 (NA) — Only 1 participant evaluable. | 16.3 (5.0) | 17.4 (NA) — Only 1 participant evaluable. | 15.8 (NA) — Only 1 participant evaluable. | 26.5 (22.6) | 25.9 (NA) — Only 1 participant evaluable. | 19.9 (29.2) |
  Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 19 | 1
  Ribociclib |  |  |  |  |  |  |  | 243 (NA) — Only 1 participant evaluable. | 161 (61.1) | 173 (NA) — Only 1 participant evaluable. | 62.4 (58.5) | 99.3 (NA) — Only 1 participant evaluable.
  Capmatinib: number analyzed (Participants) | 0 | 0 | 0 | 5 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
  Capmatinib |  |  |  | 65.9 (52.2) | 24.8 (NA) — Only 1 participant evaluable. | 45.7 (24.4) |  |  |  |  |  |
  Buparlisib: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Buparlisib | 28.2 (53.6) | 23.2 (NA) — Only 1 participant evaluable. |  |  |  |  |  |  |  |  |  |

42. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vz, ss/F) of Encorafenib, Binimetinib, Ribociclib, Capmatinib, and Buparlisib: Part II
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution is the apparent volume of distribution at steady-state.
Time Frame: as for outcome 38
Population: as for outcome 41
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 60 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 90 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Infigratinib 75 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 200 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 300 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 400 mg | Part II: Encorafenib 100 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 600 mg | Part II: Encorafenib 300 mg/Binimetinib 30 mg + Ribociclib 600 mg
Number analyzed (Participants) | 3 | 3 | 1 | 5 | 1 | 5 | 1 | 1 | 3 | 1 | 29 | 1
Liter
  Encorafenib: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 1 | 20 | 0
  Encorafenib | 268 (45.4) | 324 (69.8) | 313 (NA) — Only 1 participant evaluable. | 226 (92.9) | 91.7 (NA) — Only 1 participant evaluable. | 133 (13.5) | 177 (NA) — Only 1 participant evaluable. | 180 (NA) — Only 1 participant evaluable. | 210 (32.3) | 178 (NA) — Only 1 participant evaluable. | 99.3 (46.0) |
  Binimetinib: number analyzed (Participants) | 3 | 2 | 1 | 4 | 0 | 4 | 1 | 1 | 2 | 1 | 22 | 0
  Binimetinib | 324 (58.3) | 185 (83.4) | 82.5 (NA) — Only 1 participant evaluable. | 244 (75.9) |  | 125 (56.1) | 147 (NA) — Only 1 participant evaluable. | 86.8 (NA) — Only 1 participant evaluable. | 184 (111.8) | 406 (NA) — Only 1 participant evaluable. | 113 (48.5) |
  Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 18 | 1
  Ribociclib |  |  |  |  |  |  |  | 3160 (NA) — Only 1 participant evaluable. | 1930 (30.5) | 2660 (NA) — Only 1 participant evaluable. | 677 (65.0) | 1440 (NA) — Only 1 participant evaluable.
  Capmatinib: number analyzed (Participants) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Capmatinib |  |  |  | 190 (30.3) | 89.5 (NA) — Only 1 participant evaluable. | 233 (NA) — Only 1 participant evaluable. |  |  |  |  |  |
  Buparlisib: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Buparlisib | 604 (17.4) |  |  |  |  |  |  |  |  |  |  |

43. Secondary Outcome: Last Measurable Plasma Concentration at Steady State (Clast, ss) of Encorafenib, Binimetinib, Binimetinib Metabolite, Ribociclib, Ribociclib Metabolite, Infigratinib, Infigratinib Metabolites, Capmatinib, and Buparlisib: Part II
Time Frame: as for outcome 38
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 60 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 90 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Infigratinib 75 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 200 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 300 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 400 mg | Part II: Encorafenib 100 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 600 mg | Part II: Encorafenib 300 mg/Binimetinib 30 mg + Ribociclib 600 mg
Number analyzed (Participants) | 3 | 3 | 1 | 5 | 1 | 5 | 1 | 1 | 3 | 1 | 29 | 1
Nanogram per milliliter
  Encorafenib: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 1 | 25 | 0
  Encorafenib | 11.3 (45.3) | 25.1 (2066.8) | 6.76 (NA) — Only 1 participant evaluable. | 15.9 (315.9) | 5.20 (NA) — Only 1 participant evaluable. | 15.0 (20.9) | 10.7 (NA) — Only 1 participant evaluable. | 7.85 (NA) — Only 1 participant evaluable. | 10.8 (106.1) | 10.5 (NA) — Only 1 participant evaluable. | 33.7 (254.3) |
  Binimetinib: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 1 | 24 | 1
  Binimetinib | 44.1 (19.1) | 30.2 (59.2) | 55.8 (NA) — Only 1 participant evaluable. | 63.2 (64.0) | 17.6 (NA) — Only 1 participant evaluable. | 55.9 (54.0) | 78.3 (NA) — Only 1 participant evaluable. | 29.8 (NA) — Only 1 participant evaluable. | 23.1 (5.2) | 47.9 (NA) — Only 1 participant evaluable. | 58.7 (60.2) | 40.5 (NA) — Only 1 participant evaluable.
  Binimetinib metabolite, AR00426032: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 1 | 24 | 1
  Binimetinib metabolite, AR00426032 | 3.99 (61.8) | 2.92 (159.3) | 1.82 (NA) — Only 1 participant evaluable. | 5.57 (130.2) | 1.44 (NA) — Only 1 participant evaluable. | 4.75 (25.4) | 6.53 (NA) — Only 1 participant evaluable. | 1.08 (NA) — Only 1 participant evaluable. | 2.31 (47.8) | 3.54 (NA) — Only 1 participant evaluable. | 4.68 (92.3) | 1.56 (NA) — Only 1 participant evaluable.
  Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 26 | 1
  Ribociclib |  |  |  |  |  |  | 94.0 (NA) — Only 1 participant evaluable. | 25.6 (NA) — Only 1 participant evaluable. | 52.7 (90.4) | 34.9 (NA) — Only 1 participant evaluable. | 147 (71.8) | 91.8 (NA) — Only 1 participant evaluable.
  Ribociclib metabolite, LEQ803: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 26 | 1
  Ribociclib metabolite, LEQ803 |  |  |  |  |  |  | 84.5 (NA) — Only 1 participant evaluable. | 46.8 (NA) — Only 1 participant evaluable. | 42.5 (13.8) | 22.8 (NA) — Only 1 participant evaluable. | 73.2 (49.6) | 59.6 (NA) — Only 1 participant evaluable.
  Infigratinib: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infigratinib |  |  | 20.5 (NA) — Only 1 participant evaluable. |  |  |  |  |  |  |  |  |
  Infigratinib metabolite, BHS697: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infigratinib metabolite, BHS697 |  |  | 5.57 (NA) — Only 1 participant evaluable. |  |  |  |  |  |  |  |  |
  Infigratinib metabolite, CQM157: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infigratinib metabolite, CQM157 |  |  | 32.2 (NA) — Only 1 participant evaluable. |  |  |  |  |  |  |  |  |
  Capmatinib: number analyzed (Participants) | 0 | 0 | 0 | 5 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
  Capmatinib |  |  |  | 79.6 (103.1) | 58.1 (NA) — Only 1 participant evaluable. | 269 (68.7) |  |  |  |  |  |
  Buparlisib: number analyzed (Participants) | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Buparlisib | 41.8 (82.9) | 101 (1.4) |  |  |  |  |  |  |  |  |  |

44. Secondary Outcome: Measured Concentration at the End of a Dosing Interval at Steady State (Ctrough, ss) of Encorafenib, Binimetinib, Binimetinib Metabolite, Ribociclib, Ribociclib Metabolite, Infigratinib, Infigratinib Metabolites, Capmatinib, and Buparlisib: Part II
Time Frame: C1 D15: at the end of a dosing interval at steady-state (24 hour ± 2 hour), taken directly before next administration
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 60 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Buparlisib 90 mg | Part II: Encorafenib 450 mg/ Binimetinib 45 mg + Infigratinib 75 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 200 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 300 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Capmatinib 400 mg | Part II: Encorafenib 100 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 30 mg + Ribociclib 600 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 400 mg | Part II: Encorafenib 200 mg/ Binimetinib 45 mg + Ribociclib 600 mg | Part II: Encorafenib 300 mg/Binimetinib 30 mg + Ribociclib 600 mg
Number analyzed (Participants) | 3 | 3 | 1 | 5 | 1 | 5 | 1 | 1 | 3 | 1 | 29 | 1
Nanogram per milliliter
  Encorafenib: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 1 | 24 | 0
  Encorafenib | 11.2 (106.3) | 18.6 (159.4) | 7.74 (NA) — Only 1 participant evaluable. | 11.6 (51.3) | 7.95 (NA) — Only 1 participant evaluable. | 13.5 (35.0) | 9.28 (NA) — Only 1 participant evaluable. | 10.3 (NA) — Only 1 participant evaluable. | 7.75 (37.3) | 10.4 (NA) — Only 1 participant evaluable. | 21.7 (185.4) |
  Binimetinib: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 1 | 23 | 1
  Binimetinib | 32.0 (17.1) | 39.1 (57.4) | 33.9 (NA) — Only 1 participant evaluable. | 81.2 (47.5) | 47.3 (NA) — Only 1 participant evaluable. | 50.9 (34.4) | 54.3 (NA) — Only 1 participant evaluable. | 28.3 (NA) — Only 1 participant evaluable. | 21.1 (23.7) | 31.5 (NA) — Only 1 participant evaluable. | 51.0 (76.1) | 36.2 (NA) — Only 1 participant evaluable.
  Binimetinib metabolite, AR00426032: number analyzed (Participants) | 3 | 2 | 1 | 5 | 1 | 4 | 1 | 1 | 2 | 1 | 23 | 1
  Binimetinib metabolite, AR00426032 | 3.14 (74.5) | 3.80 (111.9) | 1.21 (NA) — Only 1 participant evaluable. | 8.22 (84.6) | 4.36 (NA) — Only 1 participant evaluable. | 5.45 (42.2) | 4.16 (NA) — Only 1 participant evaluable. | NA (NA) — Only 1 participant evaluable. | 3.81 (NA) — Only 1 participant evaluable. | 1.72 (NA) — Only 1 participant evaluable. | 4.34 (79.9) | 1.09 (NA) — Only 1 participant evaluable.
  Ribociclib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 25 | 1
  Ribociclib |  |  |  |  |  |  | 98.4 (NA) — Only 1 participant evaluable. | 28.2 (NA) — Only 1 participant evaluable. | 30.7 (24.9) | 36.4 (NA) — Only 1 participant evaluable. | 104 (54.2) | 64.7 (NA) — Only 1 participant evaluable.
  Ribociclib metabolite, LEQ803: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 25 | 1
  Ribociclib metabolite, LEQ803 |  |  |  |  |  |  | 76.0 (NA) — Only 1 participant evaluable. | 37.1 (NA) — Only 1 participant evaluable. | 32.9 (25.7) | 22.8 (NA) — Only 1 participant evaluable. | 55.1 (33.9) | 49.2 (NA) — Only 1 participant evaluable.
  Infigratinib: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infigratinib |  |  | 2.49 (NA) — Only 1 participant evaluable. |  |  |  |  |  |  |  |  |
  Infigratinib metabolite, BHS697: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infigratinib metabolite, BHS697 |  |  | 1.64 (NA) — Only 1 participant evaluable. |  |  |  |  |  |  |  |  |
  Infigratinib metabolite, CQM157: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infigratinib metabolite, CQM157 |  |  | 11.1 (NA) — Only 1 participant evaluable. |  |  |  |  |  |  |  |  |
  Capmatinib: number analyzed (Participants) | 0 | 0 | 0 | 5 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
  Capmatinib |  |  |  | 83.9 (34.0) | 71.4 (NA) — Only 1 participant evaluable. | 173 (41.2) |  |  |  |  |  |
  Buparlisib: number analyzed (Participants) | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Buparlisib | 49.7 (115.9) | 97.3 (16.2) |  |  |  |  |  |  |  |  |  |

ADVERSE EVENTS:
Time Frame: Day 1 up to 30 days after last dose (maximum treatment exposure for Part I was 403.7 weeks and for Part II was 97.0 weeks)
Description: Same event may appear as both non-SAE and SAE, but what is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. Safety set evaluated.
Arm/Group | Part I: Encorafenib + Binimetinib (Naive) | Part I: Encorafenib + Binimetinib (Non-naive) | Part II: Encorafenib + Binimetinib + Ribociclib | Part II: Encorafenib + Binimetinib + Infigratinib | Part II: Encorafenib + Binimetinib + Capmatinib | Part II: Encorafenib + Binimetinib + Buparlisib
All-Cause Mortality (participants affected / at risk) | 20/75 | 29/83 | 28/38 | 1/1 | 8/13 | 4/6
Serious Adverse Events (participants affected / at risk) | 47/75 | 37/83 | 19/38 | 0/1 | 6/13 | 4/6
Other Adverse Events (participants affected / at risk) | 75/75 | 73/83 | 33/38 | 0/1 | 11/13 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I: Encorafenib + Binimetinib (Naive) (N=75) | Part I: Encorafenib + Binimetinib (Non-naive) (N=83) | Part II: Encorafenib + Binimetinib + Ribociclib (N=38) | Part II: Encorafenib + Binimetinib + Infigratinib (N=1) | Part II: Encorafenib + Binimetinib + Capmatinib (N=13) | Part II: Encorafenib + Binimetinib + Buparlisib (N=6)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 2 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Adrenomegaly (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Exophthalmos (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Intestinal mass (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 3 | 1 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Terminal ileitis (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 6 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 4 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 4 | 1 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Chorioretinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Osteoradionecrosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Troponin T increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myopathy toxic (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0 | 0
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 3 | 2 | 0 | 0 | 0 | 0
Embolic cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hemiplegia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Paresis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part I: Encorafenib + Binimetinib (Naive) (N=75) | Part I: Encorafenib + Binimetinib (Non-naive) (N=83) | Part II: Encorafenib + Binimetinib + Ribociclib (N=38) | Part II: Encorafenib + Binimetinib + Infigratinib (N=1) | Part II: Encorafenib + Binimetinib + Capmatinib (N=13) | Part II: Encorafenib + Binimetinib + Buparlisib (N=6)
Anaemia (Blood and lymphatic system disorders) | 28 | 16 | 10 | 0 | 3 | 3
Neutropenia (Blood and lymphatic system disorders) | 6 | 2 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 5 | 0 | 0 | 0
Cataract (Eye disorders) | 4 | 4 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 5 | 5 | 0 | 0 | 0 | 0
Retinopathy (Eye disorders) | 22 | 10 | 0 | 0 | 0 | 0
Subretinal fluid (Eye disorders) | 9 | 8 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 11 | 8 | 0 | 0 | 0 | 0
Visual field defect (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 1
Asthenia (General disorders) | 3 | 6 | 0 | 0 | 0 | 0
Chills (General disorders) | 5 | 7 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 14 | 11 | 2 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 22 | 13 | 5 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 33 | 25 | 9 | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 30 | 33 | 15 | 0 | 2 | 2
Vomiting (Gastrointestinal disorders) | 15 | 22 | 10 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 5 | 3 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 31 | 27 | 6 | 0 | 1 | 0
Influenza like illness (General disorders) | 6 | 5 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 15 | 10 | 4 | 0 | 3 | 1
Pyrexia (General disorders) | 13 | 16 | 7 | 0 | 0 | 2
Conjunctivitis (Infections and infestations) | 7 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 12 | 6 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 11 | 3 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 7 | 3 | 3 | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 13 | 8 | 5 | 0 | 1 | 1
Amylase increased (Investigations) | 7 | 6 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 9 | 6 | 4 | 0 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 4 | 5 | 3 | 0 | 1 | 0
Blood creatine increased (Investigations) | 4 | 4 | 4 | 0 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 38 | 10 | 5 | 0 | 2 | 0
Blood creatinine increased (Investigations) | 7 | 10 | 4 | 0 | 2 | 0
Ejection fraction decreased (Investigations) | 6 | 6 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 7 | 2 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 12 | 8 | 2 | 0 | 2 | 1
Lipase increased (Investigations) | 11 | 7 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 7 | 5 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 4 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 14 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 | 15 | 2 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 6 | 4 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 | 7 | 3 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 6 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 9 | 1 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 8 | 5 | 4 | 0 | 0 | 0
Headache (Nervous system disorders) | 14 | 8 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 3 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 8 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 4 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 10 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 5 | 3 | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 8 | 2 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 6 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 11 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 9 | 4 | 1 | 0 | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT02159066/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT02159066/SAP_001.pdf